CLINICAL TRIAL: NCT00042289
Title: Pharmacokinetic Properties of Antiretroviral and Related Drugs During Pregnancy and Postpartum
Brief Title: Pharmacokinetic Study of Antiretroviral Drugs and Related Drugs During and After Pregnancy
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: P1026s; 10040 (Registry Identifier: DAIDS ES); IMPAACT P1026s
Record Dates: First submitted 2002-07-26; First posted 2002-08-01 (Estimated); Results first posted 2022-07-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections
Keywords: Pregnancy; Pharmacokinetics; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Cobicistat; Darunavir; elvitegravir; dolutegravir; Ritonavir; efavirenz; cobicistat mixture with darunavir; Lopinavir; Rifampin; Ethambutol; Isoniazid; Pyrazinamide; Kanamycin; Amikacin; Capreomycin; Moxifloxacin; Ofloxacin; Ethionamide; Prothionamide; terizidone; Cycloserine; Aminosalicylic Acid; bedaquiline; OPC-67683; Linezolid; pretomanid; Ethinyl Estradiol; etonogestrel; Nevirapine; amprenavir; abacavir; Indinavir; fosamprenavir; Emtricitabine; Tenofovir; tipranavir; Raltegravir Potassium; etravirine; Maraviroc; Rilpivirine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (49):
- DRV/RTV 600 or 800 or 900/100mg b.i.d. then 800 or 900/100mg b.i.d. then 600/100mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received:
  darunavir/ritonavir (DRV/RTV) 600/100 mg twice daily (b.i.d.) or 800/100 mg b.i.d. until 30 weeks gestation; then 800/100 mg b.i.d. until postpartum hospital discharge; then 600/100 mg b.i.d. after postpartum hospital discharge until 2 week postpartum PK samples are drawn.
  OR darunavir/ritonavir twice daily 600/100 mg b.i.d. or 900/100 mg b.i.d. until 30 weeks gestation; then 900/100 mg b.i.d. until postpartum hospital discharge; then 600/100 mg b.i.d. after postpartum hospital discharge until 2 week postpartum PK samples are drawn.
  Interventions: Drug: darunavir/ritonavir dosage #1; Drug: darunavir/ritonavir dosage #2; Drug: darunavir/ritonavir dosage #3
- DTG 50mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received dolutegravir (DTG) 50 mg once a day (q.d.).
  Interventions: Drug: dolutegravir
- TAF 25mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 25 mg q.d. without cobicistat or ritonavir boosting.
  Interventions: Drug: tenofovir alafenamide fumarate (TAF)
- TAF 10mg q.d. w/COBI: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 10 mg q.d. with cobicistat (COBI).
  Interventions: Drug: TAF w/cobicistat
- TAF 25mg q.d. w/COBI or RTV boosting: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 25 mg q.d. with cobicistat (COBI) or ritonavir (RTV) boosting.
  Interventions: Drug: TAF w/cobicistat or ritonavir
- EVG/COBI 150/150mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received elvitegravir/cobicistat (EVG/COBI) 150/150 mg q.d
  Interventions: Drug: elvitegravir/cobicistat
- DRV/COBI 800/150 mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received darunavir/cobicistat (DRV/COBI) 800/150 mg q.d.
  Interventions: Drug: darunavir/cobicistat
- ATV/COBI 300/150 mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received atazanavir/cobicistat (ATV/COBI) 300/150 mg q.d.
  Interventions: Drug: atazanavir/cobicistat
- EFV 600 mg q.d. (outside THA): HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received efavirenz (EFV) 600 mg q.d. (Participants outside of Thailand only)
  Interventions: Drug: efavirenz
- EFV 600mg q.d. and at least one 1st line TB drug: HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz (EFV) 600mg q.d.and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  Interventions: Drug: efavirenz; Drug: rifampicin; Drug: ethambutol; Drug: isoniazid; Drug: pyrazinamide
- LPV/RTV 800/200mg b.i.d. and at least one 1st line TB drug: HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir (LPV/RTV) 800/200mg b.i.d. and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  Interventions: Drug: lopinavir/ritonavir dosage #1; Drug: rifampicin; Drug: ethambutol; Drug: isoniazid; Drug: pyrazinamide
- No ARVs and at least two 1st line TB drugs: HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following first line TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  Interventions: Drug: rifampicin; Drug: ethambutol; Drug: isoniazid; Drug: pyrazinamide
- At least two 2nd line TB drugs w/ or w/out ARVs: HIV-infected and HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following second line TB drugs at study entry:
  Injectable agents:
  * kanamycin
  * amikacin
  * capreomycin
  Fluoroquinolones:
  * moxifloxacin
  * levofloxacin
  * ofloxacin
  Oral bacteriostatic second-line agents:
  * ethionamide/prothionamide
  * terizidone/cycloserine
  * para-aminosalicylic acid (PAS)
  Other agents:
  * high dose INH
  * bedaquiline
  * clofazamine
  * delamanid
  * linezolid
  * pretomanid
  Interventions: Drug: kanamycin; Drug: amikacin; Drug: capreomycin; Drug: moxifloxacin; Drug: levoflaxacin; Drug: ofloxacin; Drug: ethionamide/prothionamide; Drug: terizidone/cycloserine; Drug: para-aminosalicylic acid (PAS); Drug: high dose INH; Drug: bedaquiline; Drug: clofazamine; Drug: delamanid; Drug: linezolid; Drug: pretomanid
- DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d with 30-35ug EE: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received darunavir/cobicistat (DRV/COBI) 800/150 mg q.d. or atazanavir/cobicistat (ATV/COBI) 300/150 mg q.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol
  Interventions: Drug: atazanavir/cobicistat; Drug: darunavir/cobicistat; Drug: ethinyl estradiol
- DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d with ENG: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received darunavir/cobicistat (DRV/COBI) 800/150 mg q.d. or atazanavir/cobicistat (ATV/COBI) 300/150 mg q.d. postpartum and starting etonogestrel (ENG) implant
  Interventions: Drug: atazanavir/cobicistat; Drug: darunavir/cobicistat; Drug: etonogestrel implant
- EFV 600mg q.d. with 30-35ug EE: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received efavirenz (EFV) 600mg q.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol (EE)
  Interventions: Drug: efavirenz; Drug: ethinyl estradiol
- ATV/RTV/TFV 300/100/300mg q.d. with 30-35ug EE: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received atazanavir/ritonavir/tenofovir (ATV/RTV/TFV) 300/100/300 mg q.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol (EE)
  Interventions: Drug: atazanavir/ritonavir/tenofovir dosage #1; Drug: ethinyl estradiol
- NVP 200mg b.i.d: HIV-infected pregnant women ≥ 26 weeks gestation who received nevirapine (NVP) 200 mg twice a day
  Interventions: Drug: nevirapine
- APV 1200mg b.i.d: HIV-infected pregnant women ≥ 26 weeks gestation who received amprenavir (APV) 1200mg twice a day
  Interventions: Drug: amprenavir
- ABC 300mg b.i.d: HIV-infected pregnant women ≥ 20 weeks gestation who received abacavir (ABC) 300mg twice a day
  Interventions: Drug: abacavir
- LPV/RTV Arm 1: 400/100mg b.i.d: HIV-infected pregnant women ≥ 26 weeks gestation who received lopinavir/ritonavir (LPV/RTV) 400/100mg twice a day
  Interventions: Drug: lopinavir/ritonavir dosage #2
- IDV/RTV Arm 1: 800/100mg b.i.d: HIV-infected pregnant women ≥ 26 weeks gestation who received indinavir/ritonavir (IDV/RTV) 800/100 mg twice a day
  Interventions: Drug: indinavir/ritonavir dosage #1
- FPV/RTV 700/100mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received fosamprenavir/ritonavir (FPV/RTV)700/100mg twice a day
  Interventions: Drug: fosamprenavir/ritonavir
- LPV/RTV Arm 2: 400/100mg b.i.d. then 533/133mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received Kaletra (LPV/RTV) 400/100 mg twice a day until 30 weeks gestation, then 533/133 mg twice a day until results of postpartum PK evaluation were available
  Interventions: Drug: lopinavir/ritonavir dosage #2; Drug: lopinavir/ritonavir dosage #3
- ATV/RTV Arm 1: 300/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received atazanavir/ritonavir (ATV/RTV) 300/100 mg once a day
  Interventions: Drug: atazanavir/ritonavir dosage #1
- DDI 400mg or 250mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received didanosine delayed release (Videx® EC) (DDI) 400 mg once a day if weight > 60 kg; 250 mg once a day if weight < 60 kg
  Interventions: Drug: didanosine delayed release (Videx® EC)
- FTC 200mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received emtricitabine (FTC) 200 mg once a day
  Interventions: Drug: emtricitabine
- TFV 300mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir (TFV) 300 mg once a day
  Interventions: Drug: tenofovir
- TFV/ATV/RTV Arm 1: 300/300/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir/atazanavir/ritonavir (TFV/ATV/RTV) 300/300/100 mg once a day
  Interventions: Drug: atazanavir/ritonavir/tenofovir dosage #1
- NFV Arm 1: 1250mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received nelfinavir (NFV) [625 mg tablets] 1250 mg twice a day
  Interventions: Drug: nelfinavir dosage #1
- EFV 600mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz (EFV) 600 mg once a day
  Interventions: Drug: efavirenz
- TPV/RTV 500/200mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received tipranavir/ritonavir (TPV/RTV) 500/200 mg twice a day
  Interventions: Drug: tipranavir/ritonavir
- LPV/RTV Arm 3: 400/100mg b.i.d. then 600/150mg b.i.d. then 400/100mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir (LPV/RTV) tablets 400/100 mg [2 tablets] twice a day until 30 weeks gestation, then 600/150 mg [3 tablets] twice a day until postpartum hospital discharge; and 400/100 mg [2 tablets] twice a day after postpartum hospital discharge, until 2 week postpartum PK sample is drawn
  Interventions: Drug: lopinavir/ritonavir dosage #2; Drug: lopinavir/ritonavir dosage #4
- RAL 400mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received raltegravir (RAL) 400 mg twice a day
  Interventions: Drug: raltegravir
- ETR 200mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received etravirine (ETR) 200mg twice a day
  Interventions: Drug: etravirine
- MVC 150 or 300mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received maraviroc (MVC)150 mg or 300 mg twice a day
  Interventions: Drug: maraviroc
- DRV/RTV 800/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received darunavir/ritonavir (DRV/RTV) 800/100 mg once a day
  Interventions: Drug: darunavir/ritonavir dosage #4
- DRV/RTV 600/100mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received darunavir/ritonavir (DRV/RTV) 600/100 mg twice a day
  Interventions: Drug: darunavir/ritonavir dosage #1
- ATV/RTV Arm 2: 300/100mg q.d. then 400/100mg q.d. then 300/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received atazanavir/ritonavir (ATV/RTV) 300/100 mg once a day until 30 weeks gestation then 400/100 mg once a day until postpartum hospital discharge; then 300/100 mg once a day after postpartum hospital discharge until 2 week postpartum PK samples drawn
  Interventions: Drug: atazanavir/ritonavir dosage #1; Drug: atazanavir/ritonavir dosage #2
- TFV/ATV/RTV Arm 2: 300/300/100mg q.d. then 300/400/100mg q.d then 300/300/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir/atazanavir/ritonavir (TFV/ATV/RTV) 300/300/100 mg once a day until 30 weeks gestation; then 300/400/100 mg once a day until postpartum hospital discharge; then 300/300/100 mg once a day after postpartum hospital discharge until 2 week postpartum PK samples drawn
  Interventions: Drug: atazanavir/ritonavir/tenofovir dosage #1; Drug: tenofovir/atazanavir/ritonavir dosage #2
- NFV Arm 2: 1250mg b.i.d. then 1875mg b.i.d. then 1250mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received nelfinavir (NFV) [625 mg tablets] 1250 mg twice a day until 30 weeks gestation; then 1875 mg twice a day until postpartum hospital discharge; then 1250 mg twice a day after postpartum hospital discharge until 2 week postpartum PK samples drawn
  Interventions: Drug: nelfinavir dosage #1; Drug: nelfinavir dosage #2
- IDV/RTV Arm 2: 400/100mg q.d. (only THA): HIV-infected pregnant women ≥ 20 weeks gestation who received indinavir/ritonavir (IDV/RTV) 400/100 mg twice a day only to participants enrolling in Thailand
  Interventions: Drug: indinavir/ritonavir dosage #2
- LPV/RTV Arm 4: 400/100mg b.i.d. then 600/150mg b.i.d. then 400/100mg b.i.d. (only African sites): HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir (LPV/RTV, Alluvia tablets) 400/100 mg [2 tablets] twice day until 30 weeks gestation; then 600/150 mg [3 tablets] twice a day until postpartum hospital discharge; then 400/100 mg [2 tablets] twice a day after postpartum hospital discharge until 2 week postpartum PK sample drawn only to participants enrolling in Uganda
  Interventions: Drug: lopinavir/ritonavir dosage #2; Drug: lopinavir/ritonavir dosage #4
- RPV 25mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received rilpivirine (RPV) (25 mg q.d.)
  Interventions: Drug: rilpivirine
- NVP 200mg b.i.d. and RIF and at least one 1st line TB drug: HIV-infected pregnant women > 20 weeks gestation who received nevirapine (NVP) 200 mg b.i.d AND rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w. and at least one of the following drugs at study entry:
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  Interventions: Drug: ethambutol; Drug: isoniazid; Drug: pyrazinamide; Drug: nevirapine
- ATV/RTV/TFV 300/100/300mg q.d. with ENG: HIV- infected women 2-12 weeks postpartum who received atazanavir/ritonavir/tenofovir (ATV/RTV/TFV) 300/100/300 mg q.d. postpartum and starting postpartum etonogestrel (ENG) implant
  Interventions: Drug: atazanavir/ritonavir/tenofovir dosage #1; Drug: etonogestrel implant
- LPV/RTV 400/100 b.i.d. with 30-35ug EE: HIV- infected women 2-12 weeks postpartum who received lopinavir/ritonavir (LPV/RTV) 400/100 b.i.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol (EE)
  Interventions: Drug: ethinyl estradiol; Drug: lopinavir/ritonavir dosage #2
- LPV/RTV 400/100 b.i.d. with ENG: HIV- infected women 2-12 weeks postpartum who received lopinavir/ritonavir (LPV/RTV) 400/100 b.i.d. postpartum and starting postpartum etonogestrel (ENG) implant
  Interventions: Drug: etonogestrel implant; Drug: lopinavir/ritonavir dosage #2
- EFV 600mg q.d. with ENG: HIV-infected women 2-12 weeks postpartum who received efavirenz (EFV) 600mg q.d. postpartum and starting postpartum etonogestrel (ENG) implant
  Interventions: Drug: efavirenz; Drug: etonogestrel implant

INTERVENTIONS:
Drug: atazanavir/cobicistat — atazanavir/cobicistat 300/150 mg q.d.
  Groups: ATV/COBI 300/150 mg q.d.; DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d with 30-35ug EE; DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d with ENG
Drug: darunavir/ritonavir dosage #1 — darunavir/ritonavir twice daily 600/100 mg b.i.d.
  Groups: DRV/RTV 600 or 800 or 900/100mg b.i.d. then 800 or 900/100mg b.i.d. then 600/100mg b.i.d.; DRV/RTV 600/100mg b.i.d.
Drug: darunavir/ritonavir dosage #2 — darunavir/ritonavir twice daily 800/100 mg b.i.d.
  Groups: DRV/RTV 600 or 800 or 900/100mg b.i.d. then 800 or 900/100mg b.i.d. then 600/100mg b.i.d.
Drug: darunavir/ritonavir dosage #3 — darunavir/ritonavir twice daily 900/100 mg b.i.d.
  Groups: DRV/RTV 600 or 800 or 900/100mg b.i.d. then 800 or 900/100mg b.i.d. then 600/100mg b.i.d.
Drug: elvitegravir/cobicistat — elvitegravir/cobicistat 150/150 mg q.d.
  Groups: EVG/COBI 150/150mg q.d.
Drug: dolutegravir — dolutegravir 50 mg q.d.
  Groups: DTG 50mg q.d.
Drug: tenofovir alafenamide fumarate (TAF) — TAF 25 mg q.d. without cobicistat or ritonavir boosting
  Groups: TAF 25mg q.d.
Drug: TAF w/cobicistat — TAF 10 mg q.d. with cobicistat
  Groups: TAF 10mg q.d. w/COBI
Drug: TAF w/cobicistat or ritonavir — TAF 25 mg q.d. with cobicistat or ritonavir boosting
  Groups: TAF 25mg q.d. w/COBI or RTV boosting
Drug: efavirenz — efavirenz 600 mg q.d.
  Groups: EFV 600 mg q.d. (outside THA); EFV 600mg q.d.; EFV 600mg q.d. and at least one 1st line TB drug; EFV 600mg q.d. with 30-35ug EE; EFV 600mg q.d. with ENG
Drug: darunavir/cobicistat — darunavir/cobicistat 800/150 mg q.d.
  Groups: DRV/COBI 800/150 mg q.d.; DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d with 30-35ug EE; DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d with ENG
Drug: lopinavir/ritonavir dosage #1 — lopinavir/ritonavir 800/200mg b.i.d.
  Groups: LPV/RTV 800/200mg b.i.d. and at least one 1st line TB drug
Drug: atazanavir/ritonavir/tenofovir dosage #1 — atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
  Groups: ATV/RTV/TFV 300/100/300mg q.d. with 30-35ug EE; ATV/RTV/TFV 300/100/300mg q.d. with ENG; TFV/ATV/RTV Arm 1: 300/300/100mg q.d.; TFV/ATV/RTV Arm 2: 300/300/100mg q.d. then 300/400/100mg q.d then 300/300/100mg q.d.
Drug: rifampicin — rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  Groups: EFV 600mg q.d. and at least one 1st line TB drug; LPV/RTV 800/200mg b.i.d. and at least one 1st line TB drug; No ARVs and at least two 1st line TB drugs
Drug: ethambutol — ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  Groups: EFV 600mg q.d. and at least one 1st line TB drug; LPV/RTV 800/200mg b.i.d. and at least one 1st line TB drug; NVP 200mg b.i.d. and RIF and at least one 1st line TB drug; No ARVs and at least two 1st line TB drugs
Drug: isoniazid — isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  Groups: EFV 600mg q.d. and at least one 1st line TB drug; LPV/RTV 800/200mg b.i.d. and at least one 1st line TB drug; NVP 200mg b.i.d. and RIF and at least one 1st line TB drug; No ARVs and at least two 1st line TB drugs
Drug: pyrazinamide — pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  Groups: EFV 600mg q.d. and at least one 1st line TB drug; LPV/RTV 800/200mg b.i.d. and at least one 1st line TB drug; NVP 200mg b.i.d. and RIF and at least one 1st line TB drug; No ARVs and at least two 1st line TB drugs
Drug: kanamycin — kanamycin (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: amikacin — amikacin (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: capreomycin — capreomycin (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: moxifloxacin — moxifloxacin (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: levoflaxacin — levofloxacin (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: ofloxacin — ofloxacin (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: ethionamide/prothionamide — ethionamide/prothionamide (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: terizidone/cycloserine — terizidone/cycloserine (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: para-aminosalicylic acid (PAS) — para-aminosalicylic acid (PAS) (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: high dose INH — high dose INH (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: bedaquiline — bedaquiline (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: clofazamine — clofazamine (2nd TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: delamanid — delamanid (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: linezolid — linezolid (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: pretomanid — pretomanid (2nd line TB drug)
  Groups: At least two 2nd line TB drugs w/ or w/out ARVs
Drug: ethinyl estradiol — oral contraceptives formulated with 30-35 μg ethinyl estradiol
  Groups: ATV/RTV/TFV 300/100/300mg q.d. with 30-35ug EE; DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d with 30-35ug EE; EFV 600mg q.d. with 30-35ug EE; LPV/RTV 400/100 b.i.d. with 30-35ug EE
Drug: etonogestrel implant — etonogestrel implant contraceptive
  Groups: ATV/RTV/TFV 300/100/300mg q.d. with ENG; DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d with ENG; EFV 600mg q.d. with ENG; LPV/RTV 400/100 b.i.d. with ENG
Drug: nevirapine — nevirapine 200 mg twice a day
  Groups: NVP 200mg b.i.d; NVP 200mg b.i.d. and RIF and at least one 1st line TB drug
Drug: amprenavir — amprenavir 1200mg twice a day
  Groups: APV 1200mg b.i.d
Drug: abacavir — abacavir 300mg twice a day
  Groups: ABC 300mg b.i.d
Drug: lopinavir/ritonavir dosage #2 — lopinavir/ritonavir (Kaletra) 400/100mg twice a day
  Groups: LPV/RTV 400/100 b.i.d. with 30-35ug EE; LPV/RTV 400/100 b.i.d. with ENG; LPV/RTV Arm 1: 400/100mg b.i.d; LPV/RTV Arm 2: 400/100mg b.i.d. then 533/133mg b.i.d.; LPV/RTV Arm 3: 400/100mg b.i.d. then 600/150mg b.i.d. then 400/100mg b.i.d.; LPV/RTV Arm 4: 400/100mg b.i.d. then 600/150mg b.i.d. then 400/100mg b.i.d. (only African sites)
Drug: indinavir/ritonavir dosage #1 — indinavir/ritonavir 800/100mg twice a day
  Groups: IDV/RTV Arm 1: 800/100mg b.i.d
Drug: fosamprenavir/ritonavir — fosamprenavir/ritonavir 700/100 mg twice a day
  Groups: FPV/RTV 700/100mg b.i.d.
Drug: lopinavir/ritonavir dosage #3 — lopinavir/ritonavir (Kaletra) 533/133 mg twice a day
  Groups: LPV/RTV Arm 2: 400/100mg b.i.d. then 533/133mg b.i.d.
Drug: atazanavir/ritonavir dosage #1 — atazanavir/ritonavir 300/100 mg once a day
  Groups: ATV/RTV Arm 1: 300/100mg q.d.; ATV/RTV Arm 2: 300/100mg q.d. then 400/100mg q.d. then 300/100mg q.d.
Drug: didanosine delayed release (Videx® EC) — didanosine delayed release (Videx® EC) 400 mg once a day if weight > 60 kg; 250 mg once a day if weight < 60 kg
  Groups: DDI 400mg or 250mg q.d.
Drug: emtricitabine — emtricitabine 200 mg once a day
  Groups: FTC 200mg q.d.
Drug: tenofovir — tenofovir 300 mg once a day
  Groups: TFV 300mg q.d.
Drug: nelfinavir dosage #1 — nelfinavir [625 mg tablets] 1250 mg twice a day
  Groups: NFV Arm 1: 1250mg b.i.d.; NFV Arm 2: 1250mg b.i.d. then 1875mg b.i.d. then 1250mg b.i.d.
Drug: tipranavir/ritonavir — tipranavir/ritonavir 500/200 mg twice a day
  Groups: TPV/RTV 500/200mg b.i.d.
Drug: lopinavir/ritonavir dosage #4 — lopinavir/ritonavir (Kaletra) tablets 600/150 mg [3 tablets] twice a day
  Groups: LPV/RTV Arm 3: 400/100mg b.i.d. then 600/150mg b.i.d. then 400/100mg b.i.d.; LPV/RTV Arm 4: 400/100mg b.i.d. then 600/150mg b.i.d. then 400/100mg b.i.d. (only African sites)
Drug: raltegravir — raltegravir 400 mg twice a day
  Groups: RAL 400mg b.i.d.
Drug: etravirine — etravirine 200 mg twice a day
  Groups: ETR 200mg b.i.d.
Drug: maraviroc — maraviroc 150 mg or 300 mg twice a day
  Groups: MVC 150 or 300mg b.i.d.
Drug: atazanavir/ritonavir dosage #2 — atazanavir/ritonavir 400/100mg once a day
  Groups: ATV/RTV Arm 2: 300/100mg q.d. then 400/100mg q.d. then 300/100mg q.d.
Drug: tenofovir/atazanavir/ritonavir dosage #2 — tenofovir/atazanavir/ritonavir 300/400/100 mg once a day
  Groups: TFV/ATV/RTV Arm 2: 300/300/100mg q.d. then 300/400/100mg q.d then 300/300/100mg q.d.
Drug: nelfinavir dosage #2 — nelfinavir [625 mg tablets] 1875 mg twice a day
  Groups: NFV Arm 2: 1250mg b.i.d. then 1875mg b.i.d. then 1250mg b.i.d.
Drug: indinavir/ritonavir dosage #2 — indinavir/ritonavir 400/100 mg twice a day
  Groups: IDV/RTV Arm 2: 400/100mg q.d. (only THA)
Drug: rilpivirine — rilpivirine (25 mg q.d.)
  Groups: RPV 25mg q.d.
Drug: darunavir/ritonavir dosage #4 — darunavir/ritonavir once daily 800/100 mg q.d.
  Groups: DRV/RTV 800/100mg q.d.

SUMMARY:
IMPAACT P1026s is a Phase IV prospective clinical study to evaluate the pharmacokinetics (PKs) of antiretroviral (ARV) and tuberculosis (TB) medications in pregnant women and their infants. (Pharmacokinetics are the various interactions between a drug and the body.) This study also evaluated the PKs of certain ARVs in postpartum women before and after starting hormonal contraceptives. The PKs of these drugs were evaluated by measuring the amount of medicine present in blood and/or vaginal secretions.

DETAILED DESCRIPTION:
Pregnant women experience unique physiological changes that may result in clinically significant alterations in drug PKs. Unfortunately, there have been few clinical trials to study the PKs of ARV, TB, and hormonal contraceptive drugs in pregnant women. The development of appropriate dosing regimens for the HIV-infected pregnant woman is critical to the health of both mother and fetus. Overdosing may lead to maternal adverse events and increased risk of fetal toxicity, while underdosing may lead to inadequate virologic control, increased risk of developing drug resistance mutations, and a higher rate of perinatal HIV transmission. This study evaluated the PKs of ARVs used during pregnancy; the PKs of TB drugs used during pregnancy, both in women who are HIV-positive and also taking ARVs and in women who are HIV-negative and not taking ARVs; and the PKs of hormonal contraceptive medications taken along with ARVs.

P1026s is a Phase IV clinical study. Participants were not assigned to the drugs under study, but were already receiving the drugs for clinical care by prescription of their clinical care providers. They were enrolled into study arms according to the drugs they were receiving through clinical care, and if on multiple drugs of interest, were able to enroll into multiple arms simultaneously. No drugs were provided as part of this study. This observational study was added to an existing investigational new drug (IND) number because several of the drugs were studied at a higher does than the approved dose after the PK results for the approved dose were found to be inadequate.

P1026s went through 10 protocol versions, with the first and last versions of the protocol finalized in 2002 and 2016, respectively. New study arms were added and analyzed separately with each update of the protocol version. In general, there were five main groups of study arms: HIV-infected pregnant women taking ARVs without TB treatment, HIV-infected pregnant women taking ARVs with first-line TB treatment, HIV-uninfected pregnant women taking no ARVs with first-line TB treatment, HIV-infected and HIV-uninfected pregnant women with or without ARVs with second-line TB treatment for drug-resistant TB, and HIV-infected postpartum women taking ARVs and hormonal contraceptives. The primary analysis of each arm was designed and conducted as a separate single arm evaluation of the drug (or combination of drugs) of interest.

Women who were 20 0/7 weeks to 37 6/7 weeks pregnant were enrolled in this study and remained in the study for up to 12 weeks after delivery. Postpartum women were enrolled at 2 to 12 weeks after delivery and followed until 6 to 7 weeks after starting contraceptives. Infants were enrolled in-utero and followed for 16 to 24 weeks of life. At all study visits, participants underwent a medical history, a physical exam, and blood collection. At some visits, women in some arms underwent a vaginal swab. Blood collection from the mother and the detached umbilical cord occurred during delivery. Intensive PK sampling was performed at study visits during the second and third trimester of pregnancy and/or postpartum, depending on the study arm. Additional study visits may have occurred depending on the ARV drug regimen prescribed. Infant washout PK samples were collected at 2-10, 18-28, 36-72 hours after birth, and 5-9 days of life.

There are a total of 49 study arms across all versions of P1026s protocols. Out of the 49 study arms, 2 did not have PK data* [didanosine delayed release (DDI) and lopinavir/ritonavir (LPV/RTV) African sites only]; 2 never enrolled any participants [amprenavir (APV) and nevirapine/rifampicin (NVP/RIF) with at least one first line TB drug]; 9 are in the line to be tested/analyzed due to batched analysis which has to be done after the end of the study, the lengthy process of development, validation and approval (regulatory burdens), and laboratory delays related to the COVID-19 pandemic [all TB arms and all but 3 contraceptive arms (atazanavir/ritonavir/tenofovir (ATV/RTV/TFV) with etonogestrel (ENG), efavirenz (EFV) with ENG, and LPV/RTV with ENG)]; and 8 had completion dates earlier than December 26, 2007 [nevirapine (NVP), abacavir (ABC), LPV/RTV 400/100 mg twice daily (b.i.d.), LPV/RTV 400/100mg then 533/133mg b.i.d, nelfinavir (NFV), emtricitabine (FTC), indinavir/ritonavir (IDV/RTV), and tipranavir/ritonavir]. In this submission, the Results Section presents participant flow, baseline characteristics and adverse events for all study arms (except the 2 arms that never enrolled), and outcome measure results for the 28 remaining study arms that have been completed and have final results available. For study arms completed prior to December 26, 2007, refer to the study publications in the References section for outcome measures.

For arms with very low enrollment (N<3), some results throughout the record (e.g. baseline characteristics and outcome measures) were not reported in order to avoid making individual participant data identifiable.

In the Outcome Measures section, there could be multiple outcome measures for same PK parameters (e.g. AUC12) depending on different units or summary statistics used in the analyses (such as median with range vs. median with interquartile range (IQR)).

ELIGIBILITY:
Maternal Inclusion Criteria:

* Participant must belong to one of the following 5 groups:

  1. HIV-infected pregnant women greater than or equal to 20 weeks gestation NOT on TB treatment receiving one or more of the ARV drugs/drug combinations specified in the protocol
  2. HIV-infected pregnant women greater than or equal to 20 weeks gestation receiving one of the ARV drugs/drug combinations specified in the protocol and TB treatment with at least one of the TB drugs, specified in the protocol, at study entry
  3. HIV-uninfected pregnant women greater than or equal to 20 weeks gestation receiving at least two of the first-line TB drugs, specified in the protocol, at study entry
  4. HIV-infected and HIV-uninfected pregnant women greater than or equal to 20 weeks gestation receiving at least two of the second-line TB drugs, specified in the protocol, at study entry
  5. HIV-infected women 2 to 12 weeks (14 to 84 days) post-delivery receiving one of the ARV drug combinations listed in the protocol AND starting postpartum contraceptives as listed in the protocol
* The woman must be stable on the ARV drug/drug combination and/or TB drug combination for at least 2 weeks prior to PK sampling
* If a woman is receiving a specific generic ARV formulation, the protocol team has approved this formulation
* HIV-infected pregnant women must be planning to continue on current ARV regimen until postpartum PK sampling is completed. HIV-infected postpartum women on hormonal contraceptives must be planning to continue on ARV and contraceptive regimens until final PK sampling is completed
* For HIV-infected women: confirmed HIV infection, documented by positive results from two samples collected at different time points prior to study entry. More information on this criterion can be found in the protocol.
* HIV-uninfected pregnant women must have documented negative HIV antibody test during current pregnancy. Note: adequate source documentation, including the date of specimen collection, date of testing, test performed, and test result, must be available.
* Participants enrolling in the 3rd trimester must enroll by 37 6/7 weeks gestation
* Participant can provide legal informed consent per local regulations
* If a woman has completed this study and becomes pregnant again, she may re-enroll in the study only if she is enrolled in a different arm than that studied during her initial enrollment

Maternal Exclusion Criteria:

* Women on medicines known to interfere with absorption, metabolism, or clearance of the drug being evaluated (see protocol for more information). Rifampicin is permitted for women being evaluated for TB and ARV drug interactions
* If pregnant, carrying multiple fetuses
* Clinical or laboratory toxicity that, in the opinion of the site investigator, would be likely to require a change in the medicine regimen during the period of study

Infant Enrollment Criteria:

- All infants of mothers enrolled during pregnancy (meeting criteria specified above) are enrolled, in utero, immediately after maternal enrollment.

Infant Requirements for Washout Pharmacokinetic Sampling:

* Born to HIV-infected mother enrolled during pregnancy in an ARV arm (does not include infants born to HIV-uninfected mothers receiving TB drugs)
* Birth weight greater than 1000 grams
* Is NOT receiving disallowed medications described in Section 7 of the protocol
* Does not have any severe congenital malformation or other medical condition not compatible with life or that would interfere with study participation or interpretation, as judged by the site investigator
* Born after singleton delivery (not after multiple birth)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant and postpartum women from IMPAACT US and non-US sites receiving the medicines specified in the protocol as part of clinical care and infants born to those women enrolled during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 1578 (Actual)
Dates: Start 2003-06-09 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mirochnick, MD, Study Chair — Boston Medical Center
Locations (62):
- United States (39):
  - UAB Pediatric Infectious Diseases CRS, Birmingham, Alabama
  - University of California, UC San Diego CRS- Mother-Child-Adolescent HIV Program, La Jolla, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - Univ. of California San Francisco NICHD CRS, San Francisco, California
  - Harbor UCLA Medical Ctr. NICHD CRS, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Washington Hosp. Ctr. NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Emory University School of Medicine NICHD CRS, Atlanta, Georgia
  - Med. College of Georgia School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Augusta, Georgia
  - Mt. Sinai Hosp. Med. Ctr. - Chicago, Womens & Childrens HIV Program, Chicago, Illinois
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Univ. of Illinois College of Medicine at Chicago, Dept. of Peds., Chicago, Illinois
  - Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Tulane Univ. New Orleans NICHD CRS, New Orleans, Louisiana
  - Univ. of Maryland Baltimore NICHD CRS, Baltimore, Maryland
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - Children's Hosp. of Boston NICHD CRS, Boston, Massachusetts
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - Nyu Ny Nichd Crs, New York, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - Philadelphia IMPAACT Unit CRS, Philadelphia, Pennsylvania
  - Regional Med. Ctr. at Memphis, Memphis, Tennessee
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Seattle Children's Research Institute CRS, Seattle, Washington
- Hosp. General de Agudos Buenos Aires Argentina NICHD CRS, Ciudad de Buenos Aires, Buenos Aires, Argentina
- Botswana (2):
  - Gaborone CRS, Gaborone, South-East District
  - Molepolole CRS, Gaborone
- Brazil (7):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte, Minas Gerais
  - Hosp. Santa Casa Porto Alegre Brazil NICHD CRS, Porto Alegre, Rio Grande do Sul
  - Hosp. dos Servidores Rio de Janeiro NICHD CRS, Rio de Janeiro
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagao Gesteira - UFRJ NICHD CRS, Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
  - Univ. of Sao Paulo Brazil NICHD CRS, São Paulo
- Puerto Rico (2):
  - IMPAACT/ Gamma Project/ UPR Pediatric HIV/AIDS Research CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan
- South Africa (3):
  - Wits RHI Shandukani Research Centre CRS, Johannesburg, Gauteng
  - Desmond Tutu TB Centre - Stellenbosch University (DTTC-SU) CRS, Cape Town, Western Cape
  - Famcru Crs, Tygerberg, Western Cape
- Kilimanjaro Christian Medical Centre (KCMC), Moshi, Tanzania
- Thailand (7):
  - Bhumibol Adulyadej Hosp. CRS, Sai Mai, Bangkok
  - Siriraj Hospital ,Mahidol University NICHD CRS, Bangkok, Bangkoknoi
  - Phayao Provincial Hosp. CRS, T.Tom, Muang, Changwat Phayao
  - Prapokklao Hosp. CRS, Chanthaburi
  - Chiangrai Prachanukroh Hospital NICHD CRS, Chiang Mai
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai
  - Chonburi Hosp. CRS, Chon Buri

REFERENCES:
- [Background] Loutfy MR, Walmsley SL. Treatment of HIV infection in pregnant women: antiretroviral management options. Drugs. 2004;64(5):471-88. doi: 10.2165/00003495-200464050-00002. PMID 14977385
- [Background] Mirochnick M, Capparelli E. Pharmacokinetics of antiretrovirals in pregnant women. Clin Pharmacokinet. 2004;43(15):1071-87. doi: 10.2165/00003088-200443150-00002. PMID 15568888
- [Background] Rakhmanina NY, van den Anker JN, Soldin SJ. Safety and pharmacokinetics of antiretroviral therapy during pregnancy. Ther Drug Monit. 2004 Apr;26(2):110-5. doi: 10.1097/00007691-200404000-00004. PMID 15228149
- [Background] Sullivan JL. Prevention of mother-to-child transmission of HIV--what next? J Acquir Immune Defic Syndr. 2003 Sep;34 Suppl 1:S67-72. doi: 10.1097/00126334-200309011-00010. PMID 14562860
- [Result] Best BM, Mirochnick M, Capparelli EV, Stek A, Burchett SK, Holland DT, Read JS, Smith E, Hu C, Spector SA, Connor JD; PACTG P1026s Study Team. Impact of pregnancy on abacavir pharmacokinetics. AIDS. 2006 Feb 28;20(4):553-60. doi: 10.1097/01.aids.0000210609.52836.d1. PMID 16470119
- [Result] Stek AM, Mirochnick M, Capparelli E, Best BM, Hu C, Burchett SK, Elgie C, Holland DT, Smith E, Tuomala R, Cotter A, Read JS. Reduced lopinavir exposure during pregnancy. AIDS. 2006 Oct 3;20(15):1931-9. doi: 10.1097/01.aids.0000247114.43714.90. PMID 16988514
- [Result] Aweeka FT, Stek A, Best BM, Hu C, Holland D, Hermes A, Burchett SK, Read J, Mirochnick M, Capparelli EV; International Maternal Pediatric Adolescent AIDS Clinical Trials Group (IMPAACT) P1026s Protocol Team. Lopinavir protein binding in HIV-1-infected pregnant women. HIV Med. 2010 Apr;11(4):232-8. doi: 10.1111/j.1468-1293.2009.00767.x. Epub 2009 Dec 3. PMID 20002783
- [Result] Mirochnick M, Best BM, Stek AM, Capparelli EV, Hu C, Burchett SK, Rossi SS, Hawkins E, Basar M, Smith E, Read JS; IMPAACT 1026s Study Team. Atazanavir pharmacokinetics with and without tenofovir during pregnancy. J Acquir Immune Defic Syndr. 2011 Apr 15;56(5):412-9. doi: 10.1097/QAI.0b013e31820fd093. PMID 21283017
- [Result] Capparelli EV, Aweeka F, Hitti J, Stek A, Hu C, Burchett SK, Best B, Smith E, Read JS, Watts H, Nachman S, Thorpe EM Jr, Spector SA, Jimenez E, Shearer WT, Foca M, Mirochnick M; PACTG 1026S Study Team; PACTG P1022 Study Team. Chronic administration of nevirapine during pregnancy: impact of pregnancy on pharmacokinetics. HIV Med. 2008 Apr;9(4):214-20. doi: 10.1111/j.1468-1293.2008.00553.x. PMID 18366444
- [Result] Mirochnick M, Best BM, Stek AM, Capparelli E, Hu C, Burchett SK, Holland DT, Smith E, Gaddipati S, Read JS; PACTG 1026s Study Team. Lopinavir exposure with an increased dose during pregnancy. J Acquir Immune Defic Syndr. 2008 Dec 15;49(5):485-91. doi: 10.1097/QAI.0b013e318186edd0. PMID 18989231
- [Result] Read JS, Best BM, Stek AM, Hu C, Capparelli EV, Holland DT, Burchett SK, Smith ME, Sheeran EC, Shearer WT, Febo I, Mirochnick M. Pharmacokinetics of new 625 mg nelfinavir formulation during pregnancy and postpartum. HIV Med. 2008 Nov;9(10):875-82. doi: 10.1111/j.1468-1293.2008.00640.x. Epub 2008 Sep 14. PMID 18795962
- [Result] Best BM, Stek AM, Mirochnick M, Hu C, Li H, Burchett SK, Rossi SS, Smith E, Read JS, Capparelli EV; International Maternal Pediatric Adolescent AIDS Clinical Trials Group 1026s Study Team. Lopinavir tablet pharmacokinetics with an increased dose during pregnancy. J Acquir Immune Defic Syndr. 2010 Aug;54(4):381-8. doi: 10.1097/qai.0b013e3181d6c9ed. PMID 20632458
- [Result] Stek AM, Best BM, Luo W, Capparelli E, Burchett S, Hu C, Li H, Read JS, Jennings A, Barr E, Smith E, Rossi SS, Mirochnick M. Effect of pregnancy on emtricitabine pharmacokinetics. HIV Med. 2012 Apr;13(4):226-35. doi: 10.1111/j.1468-1293.2011.00965.x. Epub 2011 Nov 30. PMID 22129166
- [Result] Cressey TR, Stek A, Capparelli E, Bowonwatanuwong C, Prommas S, Sirivatanapa P, Yuthavisuthi P, Neungton C, Huo Y, Smith E, Best BM, Mirochnick M; IMPAACT P1026s Team. Efavirenz pharmacokinetics during the third trimester of pregnancy and postpartum. J Acquir Immune Defic Syndr. 2012 Mar 1;59(3):245-52. doi: 10.1097/QAI.0b013e31823ff052. PMID 22083071
- [Result] Cressey TR, Best BM, Achalapong J, Stek A, Wang J, Chotivanich N, Yuthavisuthi P, Suriyachai P, Prommas S, Shapiro DE, Watts DH, Smith E, Capparelli E, Kreitchmann R, Mirochnick M; IMPAACT P1026s team. Reduced indinavir exposure during pregnancy. Br J Clin Pharmacol. 2013 Sep;76(3):475-83. doi: 10.1111/bcp.12078. PMID 23305215
- [Result] Kreitchmann R, Best BM, Wang J, Stek A, Caparelli E, Watts DH, Smith E, Shapiro DE, Rossi S, Burchett SK, Hawkins E, Byroads M, Cressey TR, Mirochnick M. Pharmacokinetics of an increased atazanavir dose with and without tenofovir during the third trimester of pregnancy. J Acquir Immune Defic Syndr. 2013 May 1;63(1):59-66. doi: 10.1097/QAI.0b013e318289b4d2. PMID 23392467
- [Result] Watts DH, Stek A, Best BM, Wang J, Capparelli EV, Cressey TR, Aweeka F, Lizak P, Kreitchmann R, Burchett SK, Shapiro DE, Hawkins E, Smith E, Mirochnick M; IMPAACT 1026s study team. Raltegravir pharmacokinetics during pregnancy. J Acquir Immune Defic Syndr. 2014 Dec 1;67(4):375-81. doi: 10.1097/QAI.0000000000000318. PMID 25162818
- [Result] Cressey TR, Urien S, Capparelli EV, Best BM, Buranabanjasatean S, Limtrakul A, Rawangban B, Sabsanong P, Treluyer JM, Jourdain G, Stek A, Lallemant M, Mirochnick M. Impact of body weight and missed doses on lopinavir concentrations with standard and increased lopinavir/ritonavir doses during late pregnancy. J Antimicrob Chemother. 2015 Jan;70(1):217-24. doi: 10.1093/jac/dku367. Epub 2014 Sep 25. PMID 25261418
- [Result] Aweeka FT, Hu C, Huang L, Best BM, Stek A, Lizak P, Burchett SK, Read JS, Watts H, Mirochnick M, Capparelli EV; International Maternal Pediatric Adolescent AIDS Clinical Trials Group (IMPAACT) P1026s Protocol Team. Alteration in cytochrome P450 3A4 activity as measured by a urine cortisol assay in HIV-1-infected pregnant women and relationship to antiretroviral pharmacokinetics. HIV Med. 2015 Mar;16(3):176-83. doi: 10.1111/hiv.12195. Epub 2014 Nov 18. PMID 25407158
- [Result] Colbers A, Best B, Schalkwijk S, Wang J, Stek A, Hidalgo Tenorio C, Hawkins D, Taylor G, Kreitchmann R, Burchett S, Haberl A, Kabeya K, van Kasteren M, Smith E, Capparelli E, Burger D, Mirochnick M; PANNA Network and the IMPAACT 1026 Study Team. Maraviroc Pharmacokinetics in HIV-1-Infected Pregnant Women. Clin Infect Dis. 2015 Nov 15;61(10):1582-9. doi: 10.1093/cid/civ587. Epub 2015 Jul 22. PMID 26202768
- [Result] Best BM, Burchett S, Li H, Stek A, Hu C, Wang J, Hawkins E, Byroads M, Watts DH, Smith E, Fletcher CV, Capparelli EV, Mirochnick M; International Maternal Pediatric and Adolescent AIDS Clinical Trials (IMPAACT) P1026s Team. Pharmacokinetics of tenofovir during pregnancy and postpartum. HIV Med. 2015 Sep;16(8):502-11. doi: 10.1111/hiv.12252. Epub 2015 May 11. PMID 25959631
- [Result] Stek A, Best BM, Wang J, Capparelli EV, Burchett SK, Kreitchmann R, Rungruengthanakit K, Cressey TR, Mofenson LM, Smith E, Shapiro D, Mirochnick M. Pharmacokinetics of Once Versus Twice Daily Darunavir in Pregnant HIV-Infected Women. J Acquir Immune Defic Syndr. 2015 Sep 1;70(1):33-41. doi: 10.1097/QAI.0000000000000668. PMID 25950206
- [Result] Tran AH, Best BM, Stek A, Wang J, Capparelli EV, Burchett SK, Kreitchmann R, Rungruengthanakit K, George K, Cressey TR, Chakhtoura N, Smith E, Shapiro DE, Mirochnick M; IMPAACT P1026s Protocol Team. Pharmacokinetics of Rilpivirine in HIV-Infected Pregnant Women. J Acquir Immune Defic Syndr. 2016 Jul 1;72(3):289-96. doi: 10.1097/QAI.0000000000000968. PMID 26918544
- [Result] Mulligan N, Schalkwijk S, Best BM, Colbers A, Wang J, Capparelli EV, Molto J, Stek AM, Taylor G, Smith E, Hidalgo Tenorio C, Chakhtoura N, van Kasteren M, Fletcher CV, Mirochnick M, Burger D. Etravirine Pharmacokinetics in HIV-Infected Pregnant Women. Front Pharmacol. 2016 Aug 4;7:239. doi: 10.3389/fphar.2016.00239. eCollection 2016. PMID 27540363
- [Result] Mulligan N, Best BM, Wang J, Capparelli EV, Stek A, Barr E, Buschur SL, Acosta EP, Smith E, Chakhtoura N, Burchett S, Mirochnick M; IMPAACT P1026s Protocol Team. Dolutegravir pharmacokinetics in pregnant and postpartum women living with HIV. AIDS. 2018 Mar 27;32(6):729-737. doi: 10.1097/QAD.0000000000001755. PMID 29369162
- [Result] Schalkwijk S, Ter Heine R, Colbers AC, Huitema ADR, Denti P, Dooley KE, Capparelli E, Best BM, Cressey TR, Greupink R, Russel FGM, Mirochnick M, Burger DM. A Mechanism-Based Population Pharmacokinetic Analysis Assessing the Feasibility of Efavirenz Dose Reduction to 400 mg in Pregnant Women. Clin Pharmacokinet. 2018 Nov;57(11):1421-1433. doi: 10.1007/s40262-018-0642-9. PMID 29520730
- [Result] Eke AC, Chakhtoura N, Kashuba A, Best BM, Sykes C, Wang J, Stek AM, Smith E, Calabrese S, Capparelli EV, Mirochnick M; IMPAACT P1026s Protocol Team. Rilpivirine Plasma and Cervicovaginal Concentrations in Women During Pregnancy and Postpartum. J Acquir Immune Defic Syndr. 2018 Jul 1;78(3):308-313. doi: 10.1097/QAI.0000000000001677. PMID 29528944
- [Result] Momper JD, Best BM, Wang J, Capparelli EV, Stek A, Barr E, Badell ML, Acosta EP, Purswani M, Smith E, Chakhtoura N, Park K, Burchett S, Shapiro DE, Mirochnick M; IMPAACT P1026s Protocol Team. Elvitegravir/cobicistat pharmacokinetics in pregnant and postpartum women with HIV. AIDS. 2018 Nov 13;32(17):2507-2516. doi: 10.1097/QAD.0000000000001992. PMID 30134297
- [Result] Eke AC, McCormack SA, Best BM, Stek AM, Wang J, Kreitchmann R, Shapiro D, Smith E, Mofenson LM, Capparelli EV, Mirochnick M; IMPAACT P1026s Protocol Team. Pharmacokinetics of Increased Nelfinavir Plasma Concentrations in Women During Pregnancy and Postpartum. J Clin Pharmacol. 2019 Mar;59(3):386-393. doi: 10.1002/jcph.1331. Epub 2018 Oct 25. PMID 30358179
- [Result] Kreitchmann R, Schalkwijk S, Best B, Wang J, Colbers A, Stek A, Shapiro D, Cressey T, Mirochnick M, Burger D. Efavirenz pharmacokinetics during pregnancy and infant washout. Antivir Ther. 2019;24(2):95-103. doi: 10.3851/IMP3283. PMID 30530925
- [Result] Schalkwijk S, Ter Heine R, Colbers A, Capparelli E, Best BM, Cressey TR, Greupink R, Russel FGM, Molto J, Mirochnick M, Karlsson MO, Burger DM. Evaluating darunavir/ritonavir dosing regimens for HIV-positive pregnant women using semi-mechanistic pharmacokinetic modelling. J Antimicrob Chemother. 2019 May 1;74(5):1348-1356. doi: 10.1093/jac/dky567. PMID 30715324
- [Result] Liu XI, Momper JD, Rakhmanina N, van den Anker JN, Green DJ, Burckart GJ, Best BM, Mirochnick M, Capparelli EV, Dallmann A. Physiologically Based Pharmacokinetic Models to Predict Maternal Pharmacokinetics and Fetal Exposure to Emtricitabine and Acyclovir. J Clin Pharmacol. 2020 Feb;60(2):240-255. doi: 10.1002/jcph.1515. Epub 2019 Sep 6. PMID 31489678
- [Result] Eke AC, Wang J, Amin K, Shapiro DE, Stek A, Smith E, Chakhtoura N, Basar M, George K, Knapp KM, Joao EC, Rungruengthanakit K, Capparelli E, Burchett S, Mirochnick M, Best BM; P1026s Protocol Team. Fosamprenavir with Ritonavir Pharmacokinetics during Pregnancy. Antimicrob Agents Chemother. 2020 Mar 24;64(4):e02260-19. doi: 10.1128/AAC.02260-19. Print 2020 Mar 24. PMID 32015036
- [Result] Liu XI, Momper JD, Rakhmanina NY, Green DJ, Burckart GJ, Cressey TR, Mirochnick M, Best BM, van den Anker JN, Dallmann A. Prediction of Maternal and Fetal Pharmacokinetics of Dolutegravir and Raltegravir Using Physiologically Based Pharmacokinetic Modeling. Clin Pharmacokinet. 2020 Nov;59(11):1433-1450. doi: 10.1007/s40262-020-00897-9. PMID 32451908
- [Result] Brooks KM, Momper JD, Pinilla M, Stek AM, Barr E, Weinberg A, Deville JG, Febo IL, Cielo M, George K, Denson K, Rungruengthanakit K, Shapiro DE, Smith E, Chakhtoura N, Rooney JF, Haubrich R, Espina R, Capparelli EV, Mirochnick M, Best BM; IMPAACT P1026s Protocol Team. Pharmacokinetics of tenofovir alafenamide with and without cobicistat in pregnant and postpartum women living with HIV. AIDS. 2021 Mar 1;35(3):407-417. doi: 10.1097/QAD.0000000000002767. PMID 33252495
- [Result] Eke AC, Shoji K, Best BM, Momper JD, Stek AM, Cressey TR, Mirochnick M, Capparelli EV. Population Pharmacokinetics of Tenofovir in Pregnant and Postpartum Women Using Tenofovir Disoproxil Fumarate. Antimicrob Agents Chemother. 2021 Feb 17;65(3):e02168-20. doi: 10.1128/AAC.02168-20. Print 2021 Feb 17. PMID 33318014
- [Result] Momper JD, Wang J, Stek A, Shapiro DE, Scott GB, Paul ME, Febo IL, Burchett S, Smith E, Chakhtoura N, Denson K, Rungruengthanakit K, George K, Yang DZ, Capparelli EV, Mirochnick M, Best BM; IMPAACT P1026s Protocol Team. Pharmacokinetics of darunavir and cobicistat in pregnant and postpartum women with HIV. AIDS. 2021 Jul 1;35(8):1191-1199. doi: 10.1097/QAD.0000000000002857. PMID 34076612
- [Derived] Momper JD, Wang J, Stek A, Shapiro DE, Powis KM, Paul ME, Badell ML, Browning R, Chakhtoura N, Denson K, Rungruengthanakit K, George K, Capparelli EV, Mirochnick M, Best BM; IMPAACT P1026s Protocol Team. Pharmacokinetics of Atazanavir Boosted With Cobicistat in Pregnant and Postpartum Women With HIV. J Acquir Immune Defic Syndr. 2022 Mar 1;89(3):303-309. doi: 10.1097/QAI.0000000000002856. PMID 34732682
- See also: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Corrected Version 2.1 - July 2017) — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled between 9Jun2003 and 30Dec2019 at US and non-US clinical research sites and could enroll in multiple arms, simultaneously; thus, reporting groups are not mutually exclusive and totals do not reflect the number of unique participants. There were 1578 unique participants (1037 mothers and 541 infants), including 8 mothers enrolled in 3 arms, 36 mothers enrolled in 2 arms, and 24 mother-infant pairs enrolled in 2 arms. Each arm was designed as a separate single-arm evaluation.
Groups:
- DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received:
  darunavir/ritonavir twice daily 600/100 mg b.i.d. or 800/100 mg b.i.d. until 30 weeks gestation; then 800/100 mg b.i.d. until postpartum hospital discharge; then 600/100 mg b.i.d. after postpartum hospital discharge until 2 week postpartum PK samples are drawn.
  OR darunavir/ritonavir twice daily 600/100 mg b.i.d. or 900/100 mg b.i.d. until 30 weeks gestation; then 900/100 mg b.i.d. until postpartum hospital discharge; then 600/100 mg b.i.d. after postpartum hospital discharge until 2 week postpartum PK samples are drawn.
  darunavir/ritonavir dosage #1: darunavir/ritonavir twice daily 600/100 mg b.i.d.
  darunavir/ritonavir dosage #2: darunavir/ritonavir twice daily 800/100 mg b.i.d.
  darunavir/ritonavir dosage #3: darunavir/ritonavir twice daily 900/100 mg b.i.d.
- DTG 50mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received dolutegravir 50 mg q.d.
  dolutegravir: dolutegravir 50 mg q.d.
- TAF 10mg q.d. w/COBI: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 10 mg q.d. with cobicistat.
  TAF w/cobicistat: TAF 10 mg q.d. with cobicistat
- TAF 25mg q.d. w/COBI or RTV Boosting: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 25 mg q.d. with cobicistat or ritonavir boosting.
  TAF w/cobicistat or ritonavir: TAF 25 mg q.d. with cobicistat or ritonavir boosting
- EVG/COBI 150/150mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received elvitegravir/cobicistat 150/150 mg q.d
  elvitegravir/cobicistat: elvitegravir/cobicistat 150/150 mg q.d.
- DRV/COBI 800/150 mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received darunavir/cobicistat 800/150 mg q.d.
  darunavir/cobicistat: darunavir/cobicistat 800/150 mg q.d.
- ATV/COBI 300/150 mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received atazanavir/cobicistat 300/150 mg q.d.
  atazanavir/cobicistat: atazanavir/cobicistat 300/150 mg q.d.
- EFV 600 mg q.d. (Outside THA): HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received efavirenz 600 mg q.d. (Participants outside of Thailand only)
  efavirenz: efavirenz 600 mg q.d.
- EFV 600mg q.d. and at Least One 1st Line TB Drug: HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz 600mg q.d.and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  efavirenz: efavirenz 600 mg q.d.
  rifampicin: rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  ethambutol: ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  isoniazid: isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  pyrazinamide: pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
- LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug: HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir 800/200mg b.i.d. and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  lopinavir/ritonavir dosage #1: lopinavir/ritonavir 800/200mg b.i.d.
  rifampicin: rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  ethambutol: ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  isoniazid: isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  pyrazinamide: pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
- No ARVs and at Least Two 1st Line TB Drugs: HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following first line TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  rifampicin: rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  ethambutol: ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  isoniazid: isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  pyrazinamide: pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
- At Least Two 2nd Line TB Drugs w/ or w/Out ARVs: HIV-infected and HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following second line TB drugs at study entry:
  Injectable agents:
  * kanamycin
  * amikacin
  * capreomycin
  Fluoroquinolones:
  * moxifloxacin
  * levofloxacin
  * ofloxacin
  Oral bacteriostatic second-line agents:
  * ethionamide/prothionamide
  * terizidone/cycloserine
  * para-aminosalicylic acid (PAS)
  Other agents:
  * high dose INH
  * bedaquiline
  * clofazamine
  * delamanid
  * linezolid
  * pretomanid
  kanamycin: kanamycin (2nd line TB drug)
  amikacin: amikacin (2nd line TB drug)
  capreomycin: capreomycin (2nd line TB drug)
  moxifloxacin: moxifloxacin (2nd line TB drug)
  levoflaxacin: levofloxacin (2nd line TB drug)
  ofloxacin: ofloxacin (2nd line TB drug)
  ethionamide/prothionamide: ethionamide/prothionamide (2nd line TB drug)
  terizidone/cycloserine: terizidone/cycloserine (2nd line TB drug)
  para-aminosalicylic acid (PAS): para-aminosalicylic acid (PAS) (2nd line TB drug)
  high dose INH: high dose INH (2nd line TB drug)
  bedaquiline: bedaquiline (2nd line TB drug)
  clofazamine: clofazamine (2nd TB drug)
  delamanid: delamanid (2nd line TB drug)
  linezolid: linezolid (2nd line TB drug)
  pretomanid: pretomanid (2nd line TB drug)
- DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With 30-35ug EE: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received darunavir/cobicistat 800/150 mg q.d. or atazanavir/cobicistat 300/150 mg q.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol
  atazanavir/cobicistat: atazanavir/cobicistat 300/150 mg q.d.
  darunavir/cobicistat: darunavir/cobicistat 800/150 mg q.d.
  ethinyl estradiol: oral contraceptives formulated with 30-35 μg ethinyl estradiol
- DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With ENG: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received darunavir/cobicistat 800/150 mg q.d. or atazanavir/cobicistat 300/150 mg q.d. postpartum and starting etonogestrel implant
  atazanavir/cobicistat: atazanavir/cobicistat 300/150 mg q.d.
  darunavir/cobicistat: darunavir/cobicistat 800/150 mg q.d.
  etonogestrel implant: etonogestrel implant contraceptive
- EFV 600mg q.d. With 30-35ug EE: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received efavirenz 600mg q.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol
  efavirenz: efavirenz 600 mg q.d.
  ethinyl estradiol: oral contraceptives formulated with 30-35 μg ethinyl estradiol
- ATV/RTV/TFV 300/100/300mg q.d. With 30-35ug EE: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received atazanavir/ritonavir/tenofovir 300/100/300 mg q.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol
  atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
  ethinyl estradiol: oral contraceptives formulated with 30-35 μg ethinyl estradiol
- NVP 200mg b.i.d: HIV-infected pregnant women ≥ 26 weeks gestation who received nevirapine 200 mg twice a day
  nevirapine: nevirapine 200 mg twice a day
- ABC 300mg b.i.d: HIV-infected pregnant women ≥ 20 weeks gestation who received abacavir 300mg twice a day
  abacavir: abacavir 300mg twice a day
- LPV/RTV Arm 1: 400/100mg b.i.d: HIV-infected pregnant women ≥ 26 weeks gestation who received lopinavir/ritonavir (Kaletra) 400/100mg twice a day
  lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day
- IDV/RTV Arm 1: 800/100mg b.i.d: HIV-infected pregnant women ≥ 26 weeks gestation who received indinavir/ritonavir 800/100 mg twice a day
  indinavir/ritonavir dosage #1: indinavir/ritonavir 800/100mg twice a day
- FPV/RTV 700/100mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received fosamprenavir/ritonavir 700/100mg twice a day
  fosamprenavir/ritonavir: fosamprenavir/ritonavir 700/100 mg twice a day
- LPV/RTV Arm 2: 400/100mg b.i.d. Then 533/133mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received Kaletra 400/100 mg twice a day until 30 weeks gestation, then 533/133 mg twice a day until results of postpartum PK evaluation were available
  lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day
  lopinavir/ritonavir dosage #3: lopinavir/ritonavir (Kaletra) 533/133 mg twice a day
- ATV/RTV Arm 1: 300/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received atazanavir/ritonavir 300/100 mg once a day
  atazanavir/ritonavir dosage #1: atazanavir/ritonavir 300/100 mg once a day
- DDI 400mg or 250mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received didanosine delayed release (Videx® EC) 400 mg once a day if weight > 60 kg; 250 mg once a day if weight < 60 kg
  didanosine delayed release (Videx® EC): didanosine delayed release (Videx® EC) 400 mg once a day if weight > 60 kg; 250 mg once a day if weight < 60 kg
- FTC 200mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received emtricitabine 200 mg once a day
  emtricitabine: emtricitabine 200 mg once a day
- TFV 300mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir 300 mg once a day
  tenofovir: tenofovir 300 mg once a day
- TFV/ATV/RTV Arm 1: 300/300/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir/atazanavir/ritonavir 300/300/100 mg once a day
  atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
- NFV Arm 1: 1250mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received nelfinavir [625 mg tablets] 1250 mg twice a day
  nelfinavir dosage #1: nelfinavir [625 mg tablets] 1250 mg twice a day
- EFV 600mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz 600 mg once a day
  efavirenz: efavirenz 600 mg q.d.
- TPV/RTV 500/200mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received tipranavir/ritonavir 500/200 mg twice a day
  tipranavir/ritonavir: tipranavir/ritonavir 500/200 mg twice a day
- LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir (Kaletra) tablets 400/100 mg [2 tablets] twice a day until 30 weeks gestation, then 600/150 mg [3 tablets] twice a day until postpartum hospital discharge; and 400/100 mg [2 tablets] twice a day after postpartum hospital discharge, until 2 week postpartum PK sample is drawn
  lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day
  lopinavir/ritonavir dosage #4: lopinavir/ritonavir (Kaletra) tablets 600/150 mg [3 tablets] twice a day
- RAL 400mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received raltegravir 400 mg twice a day
  raltegravir: raltegravir 400 mg twice a day
- ETR 200mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received etravirine 200mg twice a day
  etravirine: etravirine 200 mg twice a day
- MVC 150 or 300mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received maraviroc 150 mg or 300 mg twice a day
  maraviroc: maraviroc 150 mg or 300 mg twice a day
- DRV/RTV 800/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received darunavir/ritonavir 800/100 mg once a day
  darunavir/ritonavir dosage #4: darunavir/ritonavir once daily 800/100 mg q.d.
- DRV/RTV 600/100mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received darunavir/ritonavir 600/100 mg twice a day
  darunavir/ritonavir dosage #1: darunavir/ritonavir twice daily 600/100 mg b.i.d.
- ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received atazanavir/ritonavir 300/100 mg once a day until 30 weeks gestation then 400/100 mg once a day until postpartum hospital discharge; then 300/100 mg once a day after postpartum hospital discharge until 2 week postpartum PK samples drawn
  atazanavir/ritonavir dosage #1: atazanavir/ritonavir 300/100 mg once a day
  atazanavir/ritonavir dosage #2: atazanavir/ritonavir 400/100mg once a day
- TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir/atazanavir/ritonavir 300/300/100 mg once a day until 30 weeks gestation; then 300/400/100 mg once a day until postpartum hospital discharge; then 300/300/100 mg once a day after postpartum hospital discharge until 2 week postpartum PK samples drawn
  atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
  tenofovir/atazanavir/ritonavir dosage #2: tenofovir/atazanavir/ritonavir 300/400/100 mg once a day
- NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received nelfinavir [625 mg tablets] 1250 mg twice a day until 30 weeks gestation; then 1875 mg twice a day until postpartum hospital discharge; then 1250 mg twice a day after postpartum hospital discharge until 2 week postpartum PK samples drawn
  nelfinavir dosage #1: nelfinavir [625 mg tablets] 1250 mg twice a day
  nelfinavir dosage #2: nelfinavir [625 mg tablets] 1875 mg twice a day
- IDV/RTV Arm 2: 400/100mg q.d. (Only THA): HIV-infected pregnant women ≥ 20 weeks gestation who received indinavir/ritonavir 400/100 mg twice a day only to participants enrolling in Thailand
  indinavir/ritonavir dosage #2: indinavir/ritonavir 400/100 mg twice a day
- LPV/RTV Arm 4: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites): HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir (Alluvia tablets) 400/100 mg [2 tablets] twice day until 30 weeks gestation; then 600/150 mg [3 tablets] twice a day until postpartum hospital discharge; then 400/100 mg [2 tablets] twice a day after postpartum hospital discharge until 2 week postpartum PK sample drawn only to participants enrolling in Uganda
  lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day
  lopinavir/ritonavir dosage #4: lopinavir/ritonavir (Kaletra) tablets 600/150 mg [3 tablets] twice a day
- RPV 25mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received rilpivirine (25 mg q.d.)
  rilpivirine: rilpivirine (25 mg q.d.)
- ATV/RTV/TFV 300/100/300mg q.d. With ENG: HIV- infected women 2-12 weeks postpartum who received atazanavir/ritonavir/tenofovir 300/100/300 mg q.d. postpartum and starting postpartum etonogestrel implant
  atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
  etonogestrel implant: etonogestrel implant contraceptive
- LPV/RTV 400/100 b.i.d. With 30-35ug EE: HIV- infected women 2-12 weeks postpartum who received lopinavir/ritonavir 400/100 b.i.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol
  ethinyl estradiol: oral contraceptives formulated with 30-35 μg ethinyl estradiol
  lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day
- LPV/RTV 400/100 b.i.d. With ENG: HIV- infected women 2-12 weeks postpartum who received lopinavir/ritonavir 400/100 b.i.d. postpartum and starting postpartum etonogestrel implant
  etonogestrel implant: etonogestrel implant contraceptive
  lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day
- EFV 600mg q.d. With ENG: HIV-infected women 2-12 weeks postpartum who received efavirenz 600mg q.d. postpartum and starting postpartum etonogestrel implant
  efavirenz: efavirenz 600 mg q.d.
  etonogestrel implant: etonogestrel implant contraceptive
Period: Overall Study
Arm/Group | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. | DTG 50mg q.d. | TAF 25mg q.d. | TAF 10mg q.d. w/COBI | TAF 25mg q.d. w/COBI or RTV Boosting | EVG/COBI 150/150mg q.d. | DRV/COBI 800/150 mg q.d. | ATV/COBI 300/150 mg q.d. | EFV 600 mg q.d. (Outside THA) | EFV 600mg q.d. and at Least One 1st Line TB Drug | LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug | No ARVs and at Least Two 1st Line TB Drugs | At Least Two 2nd Line TB Drugs w/ or w/Out ARVs | DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With 30-35ug EE | DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With ENG | EFV 600mg q.d. With 30-35ug EE | ATV/RTV/TFV 300/100/300mg q.d. With 30-35ug EE | NVP 200mg b.i.d | ABC 300mg b.i.d | LPV/RTV Arm 1: 400/100mg b.i.d | IDV/RTV Arm 1: 800/100mg b.i.d | FPV/RTV 700/100mg b.i.d. | LPV/RTV Arm 2: 400/100mg b.i.d. Then 533/133mg b.i.d. | ATV/RTV Arm 1: 300/100mg q.d. | DDI 400mg or 250mg q.d. | FTC 200mg q.d. | TFV 300mg q.d. | TFV/ATV/RTV Arm 1: 300/300/100mg q.d. | NFV Arm 1: 1250mg b.i.d. | EFV 600mg q.d. | TPV/RTV 500/200mg b.i.d. | LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. | RAL 400mg b.i.d. | ETR 200mg b.i.d. | MVC 150 or 300mg b.i.d. | DRV/RTV 800/100mg q.d. | DRV/RTV 600/100mg b.i.d. | ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. | TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. | NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d. | IDV/RTV Arm 2: 400/100mg q.d. (Only THA) | LPV/RTV Arm 4: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites) | RPV 25mg q.d. | ATV/RTV/TFV 300/100/300mg q.d. With ENG | LPV/RTV 400/100 b.i.d. With 30-35ug EE | LPV/RTV 400/100 b.i.d. With ENG | EFV 600mg q.d. With ENG
Started | 26 | 30 | 27 | 33 | 29 | 31 | 28 | 12 | 27 | 24 | 2 | 27 | 13 | 2 | 6 | 29 | 28 | 12 | 26 | 17 | 1 | 30 | 29 | 22 | 18 | 21 | 28 | 25 | 29 | 25 | 1 | 35 | 43 | 16 | 12 | 32 | 36 | 38 | 35 | 18 | 26 | 25 | 32 | 25 | 27 | 27 | 28
Infant Started | 25 | 30 | 27 | 32 | 28 | 31 | 27 | 12 | 26 | 23 | 2 | 27 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 22 | 4 | 5 | 0 | 21 | 0 | 21 | 0 | 0 | 6 | 6 | 4 | 0 | 9 | 38 | 35 | 0 | 26 | 25 | 30 | 0 | 0 | 0 | 0
Infant Completed | 21 | 28 | 27 | 29 | 26 | 25 | 26 | 10 | 25 | 20 | 2 | 24 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 20 | 3 | 5 | 0 | 20 | 0 | 21 | 0 | 0 | 6 | 4 | 4 | 0 | 8 | 35 | 34 | 0 | 26 | 21 | 27 | 0 | 0 | 0 | 0
Completed | 19 | 29 | 27 | 25 | 26 | 25 | 22 | 10 | 26 | 23 | 2 | 27 | 11 | 2 | 6 | 28 | 27 | 12 | 18 | 13 | 1 | 26 | 27 | 17 | 17 | 20 | 20 | 22 | 21 | 25 | 0 | 26 | 38 | 10 | 10 | 27 | 32 | 36 | 33 | 13 | 26 | 22 | 25 | 22 | 27 | 26 | 27
Not Completed | 7 | 1 | 0 | 8 | 3 | 6 | 6 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 8 | 4 | 0 | 4 | 2 | 5 | 1 | 1 | 8 | 3 | 8 | 0 | 1 | 9 | 5 | 6 | 2 | 5 | 4 | 2 | 2 | 5 | 0 | 3 | 7 | 3 | 0 | 1 | 1
Not completed — Lost to Follow-up | 3 | 0 | 0 | 1 | 3 | 3 | 6 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 5 | 0 | 2 | 2 | 0 | 0 | 1 | 0
Not completed — Other reason | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Severe debilitation, unable to continue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site closed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant not willing to adhere to requirements | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is all mothers enrolled. Each study arm was designed as a separate single-arm evaluation. Participants were able to enroll in multiple arms, simultaneously; thus, the reporting groups are not mutually exclusive and totals do not represent the number of unique participants. There were 1037 unique mothers, including 8 who enrolled in 3 arms and 60 who enrolled in 2 arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. | DTG 50mg q.d. | TAF 25mg q.d. | TAF 10mg q.d. w/COBI | TAF 25mg q.d. w/COBI or RTV Boosting | EVG/COBI 150/150mg q.d. | DRV/COBI 800/150 mg q.d. | ATV/COBI 300/150 mg q.d. | EFV 600 mg q.d. (Outside THA) | EFV 600mg q.d. and at Least One 1st Line TB Drug | LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug | No ARVs and at Least Two 1st Line TB Drugs | At Least Two 2nd Line TB Drugs w/ or w/Out ARVs | DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With 30-35ug EE | DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With ENG | EFV 600mg q.d. With 30-35ug EE | ATV/RTV/TFV 300/100/300mg q.d. With 30-35ug EE | NVP 200mg b.i.d | ABC 300mg b.i.d | LPV/RTV Arm 1: 400/100mg b.i.d | IDV/RTV Arm 1: 800/100mg b.i.d | FPV/RTV 700/100mg b.i.d. | LPV/RTV Arm 2: 400/100mg b.i.d. Then 533/133mg b.i.d. | ATV/RTV Arm 1: 300/100mg q.d. | DDI 400mg or 250mg q.d. | FTC 200mg q.d. | TFV 300mg q.d. | TFV/ATV/RTV Arm 1: 300/300/100mg q.d. | NFV Arm 1: 1250mg b.i.d. | EFV 600mg q.d. | TPV/RTV 500/200mg b.i.d. | LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. | RAL 400mg b.i.d. | ETR 200mg b.i.d. | MVC 150 or 300mg b.i.d. | DRV/RTV 800/100mg q.d. | DRV/RTV 600/100mg b.i.d. | ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. | TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. | NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d. | IDV/RTV Arm 2: 400/100mg q.d. (Only THA) | LPV/RTV Arm 4: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites) | RPV 25mg q.d. | ATV/RTV/TFV 300/100/300mg q.d. With ENG | LPV/RTV 400/100 b.i.d. With 30-35ug EE | LPV/RTV 400/100 b.i.d. With ENG | EFV 600mg q.d. With ENG | Total
Number analyzed (Participants) | 26 | 30 | 27 | 33 | 29 | 31 | 28 | 12 | 27 | 24 | 2 | 27 | 13 | 2 | 6 | 29 | 28 | 12 | 26 | 17 | 1 | 30 | 29 | 22 | 18 | 21 | 28 | 25 | 29 | 25 | 1 | 35 | 43 | 16 | 12 | 32 | 36 | 38 | 35 | 18 | 26 | 25 | 32 | 25 | 27 | 27 | 28 | 1113
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Reporting groups are not mutually exclusive. As such, the numbers in the Total column generated automatically by ClinicalTrials.gov count participants (8 mothers who enrolled in 3 arms and 60 mothers who enrolled in 2 arms) multiple times. For arms with very low enrollment (N<3 participants), no aggregate data are available. Individual participant ages are not entered to avoid making participants identifiable; results from these arms are excluded. Results are shown for N=1032 mothers.
  years
    number analyzed (Participants) | 26 | 30 | 27 | 33 | 29 | 31 | 28 | 12 | 27 | 24 | 0 | 27 | 13 | 0 | 6 | 29 | 28 | 12 | 26 | 17 | 0 | 30 | 29 | 22 | 18 | 21 | 28 | 25 | 29 | 25 | 0 | 35 | 43 | 16 | 12 | 32 | 36 | 38 | 35 | 18 | 26 | 25 | 32 | 25 | 27 | 27 | 28 | 1107
    (all) | 28.8 [21.3 to 34.1] | 31.8 [26.7 to 33.8] | 29.3 [24.0 to 35.1] | 33.6 [26.6 to 35.2] | 30.8 [25.3 to 36.1] | 32.1 [26.3 to 34.6] | 27.7 [22.7 to 31.8] | 33.1 [29.3 to 38.4] | 30.6 [28.2 to 34.9] | 31.4 [26.3 to 34.0] |  | 25.9 [22.0 to 30.2] | 32.5 [28.5 to 34.3] |  | 33.2 [26.4 to 35.2] | 27.1 [22.7 to 34.6] | 32.0 [27.6 to 33.6] | 29.5 [24.6 to 34.2] | 28.4 [24.8 to 33.5] | 31.4 [28.1 to 33.5] |  | 30.7 [25.4 to 34.0] | 31.8 [27.6 to 35.2] | 31.1 [23.8 to 35.2] | 28.7 [21.3 to 36.9] | 29.6 [21.9 to 32.2] | 30.2 [25.8 to 33.8] | 31.0 [26.8 to 34.2] | 28.7 [22.9 to 34.5] | 29.3 [25.2 to 32.9] |  | 30.4 [27.1 to 34.9] | 30.5 [24.8 to 34.5] | 25.5 [20.7 to 28.1] | 23.8 [21.4 to 25.1] | 27.6 [22.8 to 33.0] | 27.0 [22.0 to 34.3] | 31.0 [27.0 to 35.2] | 26.9 [23.2 to 33.7] | 28.6 [24.0 to 32.1] | 30.4 [24.0 to 33.2] | 29.0 [23.5 to 31.1] | 26.7 [23.9 to 31.0] | 26.9 [21.8 to 31.6] | 29.4 [24.1 to 35.8] | 26.9 [22.4 to 31.5] | 24.3 [21.7 to 30.8] | 29.4 [24.3 to 33.9]
Sex: Female, Male [Count of Participants; unit: Participants] — Reporting groups are not mutually exclusive. As such, the numbers in the Total column generated automatically by ClinicalTrials.gov count participants (8 mothers who enrolled in 3 arms and 60 mothers who enrolled in 2 arms) multiple times.
  Participants
    Female | 26 | 30 | 27 | 33 | 29 | 31 | 28 | 12 | 27 | 24 | 2 | 27 | 13 | 2 | 6 | 29 | 28 | 12 | 26 | 17 | 1 | 30 | 29 | 22 | 18 | 21 | 28 | 25 | 29 | 25 | 1 | 35 | 43 | 16 | 12 | 32 | 36 | 38 | 35 | 18 | 26 | 25 | 32 | 25 | 27 | 27 | 28 | 1113
    Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Reporting groups are not mutually exclusive. As such, the numbers in the Total column generated automatically by ClinicalTrials.gov count participants (8 mothers who enrolled in 3 arms and 60 mothers who enrolled in 2 arms) multiple times. For arms with very low enrollment (N<3 participants), no aggregate data are available. Individual races/ethnicities are not entered to avoid making participants identifiable; results from these arms are excluded. Results are shown for N=1032 mothers.
  Participants
    number analyzed (Participants) | 26 | 30 | 27 | 33 | 29 | 31 | 28 | 12 | 27 | 24 | 0 | 27 | 12 | 0 | 6 | 29 | 28 | 11 | 26 | 16 | 0 | 30 | 29 | 22 | 17 | 21 | 28 | 24 | 29 | 25 | 0 | 35 | 43 | 16 | 12 | 32 | 36 | 38 | 35 | 18 | 26 | 25 | 32 | 25 | 27 | 27 | 28 | 1102
    White Non-Hispanic | 0 | 3 | 4 | 3 | 1 | 3 | 0 | 2 | 0 | 0 |  | 0 | 0 |  | 0 | 0 | 1 | 2 | 4 | 1 |  | 1 | 7 | 1 | 1 | 6 | 8 | 4 | 1 | 0 |  | 6 | 3 | 0 | 0 | 2 | 4 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 74
    Black Non-Hispanic | 13 | 21 | 8 | 20 | 14 | 22 | 18 | 6 | 12 | 21 |  | 14 | 12 |  | 3 | 1 | 6 | 5 | 14 | 7 |  | 13 | 10 | 14 | 5 | 6 | 9 | 12 | 17 | 1 |  | 7 | 21 | 7 | 4 | 18 | 12 | 5 | 15 | 10 | 0 | 25 | 18 | 6 | 3 | 1 | 0 | 456
    Hispanic (Regardless of Race) | 12 | 4 | 14 | 10 | 13 | 5 | 10 | 2 | 15 | 1 |  | 4 | 0 |  | 3 | 16 | 20 | 4 | 7 | 7 |  | 15 | 11 | 7 | 11 | 7 | 10 | 7 | 11 | 2 |  | 22 | 18 | 9 | 7 | 11 | 15 | 16 | 16 | 6 | 0 | 0 | 12 | 19 | 24 | 26 | 20 | 449
    Asian, Pacific Islander | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 2 |  | 9 | 0 |  | 0 | 12 | 1 | 0 | 1 | 1 |  | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 21 |  | 0 | 0 | 0 | 0 | 0 | 4 | 17 | 0 | 0 | 26 | 0 | 1 | 0 | 0 | 0 | 8 | 112
    American Indian, Alaskan Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    More Than One Race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |  | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: PK Parameter: Area Under the Curve From 0 to 12 Hours (AUC12) With Median (IQR) for ARVs and TB Drugs
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. AUC12 (area under the curve from 0 to 12 hours) were determined using the linear trapezoidal rule.
Time Frame: Measured in 2nd trimester (20-26 wks gestation), 3rd trimester (30-38 wks gestation), and either 2-3 wks, 2-8 wks, or 6-12 wks postpartum depending on study arm. Blood samples were drawn pre-dose and at 1, 2, 4, 6, 8, and 12 hrs post dosing.
Population: All mothers with intensive pharmacokinetic (PK) results taking the dose under study at that time period (2nd trimester, 3rd trimester or postpartum). Because participants could enter the study at different time period per the study design, they are not expected to have results at every time period.
Measure: Median (Inter-Quartile Range); unit: mg*hour/L
Groups:
- DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received:
  darunavir/ritonavir (DRV/RTV) twice daily 600/100 mg b.i.d. or 800/100 mg b.i.d. until 30 weeks gestation; then 800/100 mg b.i.d. until postpartum hospital discharge; then 600/100 mg b.i.d. after postpartum hospital discharge until 2 week postpartum PK samples are drawn.
  OR darunavir/ritonavir twice daily 600/100 mg b.i.d. or 900/100 mg b.i.d. until 30 weeks gestation; then 900/100 mg b.i.d. until postpartum hospital discharge; then 600/100 mg b.i.d. after postpartum hospital discharge until 2 week postpartum PK samples are drawn.
  darunavir/ritonavir dosage #1: darunavir/ritonavir twice daily 600/100 mg b.i.d.
  darunavir/ritonavir dosage #2: darunavir/ritonavir twice daily 800/100 mg b.i.d.
  darunavir/ritonavir dosage #3: darunavir/ritonavir twice daily 900/100 mg b.i.d.
Arm/Group | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. | FPV/RTV 700/100mg b.i.d. | DRV/RTV 600/100mg b.i.d. | NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d.
Number analyzed (Participants) | 24 | 29 | 34 | 18
mg*hour/L
  2nd Trimester: number analyzed (Participants) | 9 | 8 | 13 | 18
  2nd Trimester | 55.1 [46.4 to 57.7] | 43.50 [38.50 to 50.40] | 45.8 [36.1 to 53.4] | NA [NA to NA] — PK parameters not calculated for the 2nd trimester
  3rd Trimester: number analyzed (Participants) | 24 | 28 | 34 | 18
  3rd Trimester | 51.8 [41.2 to 57.7] | 32.15 [21.45 to 39.70] | 45.9 [29.3 to 52.5] | 34.2 [27.2 to 46.9]
  Postpartum: number analyzed (Participants) | 24 | 22 | 27 | 16
  Postpartum | 79.6 [66.6 to 103.0] | 51.60 [45.20 to 59.60] | 61.7 [49.7 to 80.9] | 33.5 [28.6 to 43.5]
Statistical Analysis 1: Comparison: DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d; Test type: Superiority; p = 0.055, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.62, 90% CI 2-sided [0.44 to 0.88]
Statistical Analysis 2: Comparison: DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d; Test type: Superiority; p < 0.001, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.64, 90% CI 2-sided [0.55 to 0.73]
Statistical Analysis 3: Comparison: FPV/RTV 700/100mg b.i.d; Test type: Superiority; p = 0.22, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.68, 90% CI 2-sided [0.44 to 1.04]
Statistical Analysis 4: Comparison: FPV/RTV 700/100mg b.i.d; Test type: Superiority; p < 0.001, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.60, 90% CI 2-sided [0.49 to 0.72]
Statistical Analysis 5: Comparison: DRV/RTV 600/100mg b.i.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.76, 90% CI 2-sided [0.64 to 0.89]
Statistical Analysis 6: Comparison: DRV/RTV 600/100mg b.i.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.71, 90% CI 2-sided [0.57 to 0.88]
Statistical Analysis 7: Comparison: NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d; Test type: Superiority; p = 0.78, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.98, 90% CI 2-sided [0.71 to 1.35]

2. Primary Outcome: PK Parameter: Area Under the Curve From 0 to 12 Hours (AUC12) With Median (Range) for ARVs and TB Drugs
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: mg*hour/L
Arm/Group | LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. | RAL 400mg b.i.d. | ETR 200mg b.i.d. | IDV/RTV Arm 2: 400/100mg q.d. (Only THA)
Number analyzed (Participants) | 33 | 42 | 15 | 26
mg*hour/L
  2nd Trimester: number analyzed (Participants) | 11 | 16 | 5 | 13
  2nd Trimester | 72 [47 to 93] | 6.6 [2.1 to 18.5] | 4.5 [3.4 to 10.7] | 14.9 [10.4 to 38.7]
  3rd Trimester: number analyzed (Participants) | 33 | 41 | 13 | 25
  3rd Trimester | 96 [43 to 198] | 5.4 [1.4 to 35.6] | 8.3 [2.7 to 31.0] | 16.1 [7.5 to 39.9]
  Postpartum: number analyzed (Participants) | 27 | 38 | 8 | 26
  Postpartum | 133 [66 to 237] | 11.6 [1.6 to 39.9] | 5.3 [2.1 to 16.4] | 27.1 [18.6 to 44.7]
Statistical Analysis 1: Comparison: LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.51, 90% CI 2-sided [0.42 to 0.63]
Statistical Analysis 2: Comparison: LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.73, 90% CI 2-sided [0.63 to 0.84]
Statistical Analysis 3: Comparison: RAL 400mg b.i.d; Test type: Superiority; p = 0.03, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.58, 90% CI 2-sided [0.34 to 0.98]
Statistical Analysis 4: Comparison: RAL 400mg b.i.d; Test type: Superiority; p = 0.001, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.67, 90% CI 2-sided [0.51 to 0.89]
Statistical Analysis 5: Comparison: ETR 200mg b.i.d; Test type: Superiority; p = 0.0684, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum [Note: Comparison of 2nd Trimester vs. Postpartum was not done due to low sample size.]; Geometric mean ratio = 1.34
Statistical Analysis 6: Comparison: IDV/RTV Arm 2: 400/100mg q.d. (Only THA); Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.58, 90% CI 2-sided [0.49 to 0.68]
Statistical Analysis 7: Comparison: IDV/RTV Arm 2: 400/100mg q.d. (Only THA); Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.60, 90% CI 2-sided [0.53 to 0.68]

3. Primary Outcome: PK Parameter: Area Under the Curve From 0 to 12 Hours (AUC12) With Geometric Mean (95% CI) for ARVs and TB Drugs
Description: Measured in 2nd trimester (20-26 wks gestation), 3rd trimester (30-38 wks gestation), and either 2-3 wks, 2-8 wks, or 6-12 wks postpartum depending on study arm. Blood samples were drawn pre-dose and at 1, 2, 4, 6, 8, and 12 hrs post dosing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hour/mL
Arm/Group | MVC 150 or 300mg b.i.d.
Number analyzed (Participants) | 18
ng*hour/mL
  2nd Trimester | NA [NA to NA] — PK parameters not calculated for the 2nd trimester
  3rd Trimester: number analyzed (Participants) | 12
  3rd Trimester | 2717 [2038 to 3622]
  Postpartum: number analyzed (Participants) | 10
  Postpartum | 3645 [2429 to 5469]
Statistical Analysis 1: Comparison: MVC 150 or 300mg b.i.d; Test type: Superiority; p = 0.008, t-test, 2 sided — 3rd Trimester vs. Postpartum; Paired sample t-test on natural log-transformed PK parameter; Geometric mean ratio = 0.72, 90% CI 2-sided [0.60 to 0.88]

4. Primary Outcome: PK Parameter: Area Under the Curve From 0 to 24 Hours (AUC24) With Median (IQR) for ARVs and TB Drugs
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. AUC24 (area under the curve from 0 to 24 hours) were determined using the linear trapezoidal rule.
Time Frame: Measured at 2nd trimester (20-26 wks gestation), 3rd trimester (30-38 wks gestation), and either 2-3 wks, 2-8 wks or 6-12 wks postpartum depending on study arm. Blood samples were drawn pre-dose and at 1, 2, 4, 6, 8, 12 and 24 hours post dosing.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg*hour/L
Groups:
- DTG 50mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received dolutegravir (DTG) 50 mg q.d.
  dolutegravir: dolutegravir 50 mg q.d.
Arm/Group | DTG 50mg q.d. | TAF 25mg q.d. | TAF 10mg q.d. w/COBI | TAF 25mg q.d. w/COBI or RTV Boosting | EVG/COBI 150/150mg q.d. | DRV/COBI 800/150 mg q.d. | ATV/COBI 300/150 mg q.d. | EFV 600 mg q.d. (Outside THA) | ATV/RTV Arm 1: 300/100mg q.d. | TFV 300mg q.d. | TFV/ATV/RTV Arm 1: 300/300/100mg q.d. | DRV/RTV 800/100mg q.d. | ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. | TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d.
Number analyzed (Participants) | 29 | 27 | 31 | 29 | 30 | 29 | 11 | 42 | 18 | 37 | 20 | 32 | 37 | 35
mg*hour/L
  2nd Trimester: number analyzed (Participants) | 15 | 15 | 17 | 12 | 17 | 16 | 6 | 15 | 1 | 4 | 4 | 15 | 14 | 17
  2nd Trimester | 47.6 [33.4 to 63.7] | 0.171 [0.147 to 0.217] | 0.197 [0.145 to 0.354] | 0.181 [0.133 to 0.549] | 15.3 [11.9 to 19.0] | 50.00 [27.032 to 58.90] | 25.33 [20.95 to 27.32] | 47.30 [40.10 to 79.70] | 88.2 [NA to NA] — IQR could not be estimated since only one AUC was calculated | 1.9 [1.7 to 2.5] | 14.5 [11.3 to 21.0] | 64.6 [35.9 to 72.3] | 30.6 [19.9 to 39.0] | 26.2 [19.9 to 38.4]
  3rd Trimester: number analyzed (Participants) | 28 | 27 | 26 | 27 | 26 | 26 | 8 | 42 | 18 | 37 | 20 | 30 | 37 | 32
  3rd Trimester | 49.2 [36.4 to 62.0] | 0.212 [0.153 to 0.290] | 0.206 [0.158 to 0.284] | 0.257 [0.173 to 0.445] | 14.0 [9.1 to 18.8] | 42.05 [26.83 to 50.50] | 18.85 [11.90 to 31.48] | 60.02 [42.96 to 85.40] | 41.9 [27.4 to 60.8] | 2.4 [1.9 to 3.1] | 28.8 [15.4 to 34.5] | 63.5 [46.0 to 75.2] | 45.7 [30.8 to 57.3] | 37.7 [25.7 to 44.4]
  Postpartum: number analyzed (Participants) | 22 | 25 | 23 | 21 | 25 | 19 | 9 | 40 | 13 | 32 | 19 | 23 | 34 | 34
  Postpartum | 65.0 [47.8 to 88.4] | 0.271 [0.178 to 0.561] | 0.216 [0.164 to 0.457] | 0.283 [0.161 to 0.507] | 21.0 [13.5 to 32.8] | 95.55 [67.20 to 118.95] | 36.20 [24.09 to 46.14] | 62.70 [43.75 to 87.51] | 57.9 [47.1 to 64.8] | 3.0 [2.2 to 3.7] | 39.6 [21.0 to 54.9] | 103.9 [85.9 to 135.7] | 48.8 [34.9 to 67.5] | 58.7 [41.4 to 80.5]
Statistical Analysis 1: Comparison: DTG 50mg q.d; Test type: Superiority; p = 0.002, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.63, 90% CI 2-sided [0.52 to 0.75]
Statistical Analysis 2: Comparison: DTG 50mg q.d; Test type: Superiority; p = 0.0003, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.71, 90% CI 2-sided [0.63 to 0.81]
Statistical Analysis 3: Comparison: TAF 25mg q.d; Test type: Superiority; p = 0.09, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.57, 90% CI 2-sided [0.34 to 0.98]
Statistical Analysis 4: Comparison: TAF 25mg q.d; Test type: Superiority; p = 0.004, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.67, 90% CI 2-sided [0.54 to 0.82]
Statistical Analysis 5: Comparison: TAF 10mg q.d. w/COBI; Test type: Superiority; p = 0.27, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.79, 90% CI 2-sided [0.50 to 1.27]
Statistical Analysis 6: Comparison: TAF 10mg q.d. w/COBI; Test type: Superiority; p = 0.70, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.86, 90% CI 2-sided [0.66 to 1.12]
Statistical Analysis 7: Comparison: TAF 25mg q.d. w/COBI or RTV Boosting; Test type: Superiority; p = 0.46, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.62, 90% CI 2-sided [0.29 to 1.34]
Statistical Analysis 8: Comparison: TAF 25mg q.d. w/COBI or RTV Boosting; Test type: Superiority; p = 0.50, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.94, 90% CI 2-sided [0.63 to 1.39]
Statistical Analysis 9: Comparison: EVG/COBI 150/150mg q.d; Test type: Superiority; p < 0.10, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.76, 90% CI 2-sided [0.57 to 1.0]
Statistical Analysis 10: Comparison: EVG/COBI 150/150mg q.d; Test type: Superiority; p < 0.10, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.56, 90% CI 2-sided [0.42 to 0.73]
Statistical Analysis 11: Comparison: DRV/COBI 800/150 mg q.d; Test type: Superiority; p < 0.10, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.47, 90% CI 2-sided [0.33 to 0.68]
Statistical Analysis 12: Comparison: DRV/COBI 800/150 mg q.d; Test type: Superiority; p < 0.10, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.44, 90% CI 2-sided [0.36 to 0.54]
Statistical Analysis 13: Comparison: ATV/COBI 300/150 mg q.d; Test type: Superiority; p = 0.1875, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.74, 90% CI 2-sided [0.53 to 1.04]
Statistical Analysis 14: Comparison: ATV/COBI 300/150 mg q.d; Test type: Superiority; p = 0.1563, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.46, 90% CI 2-sided [0.19 to 1.11]
Statistical Analysis 15: Comparison: EFV 600 mg q.d. (Outside THA); Test type: Superiority; p = 0.241, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.94, 90% CI 2-sided [0.85 to 1.03]
Statistical Analysis 16: Comparison: EFV 600 mg q.d. (Outside THA); Test type: Superiority; p = 0.837, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 1.09, 90% CI 2-sided [0.90 to 1.32]
Statistical Analysis 17: Comparison: ATV/RTV Arm 1: 300/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum [Note: Comparison of 2nd Trimester vs. Postpartum was not done due to low sample size.]; Geometric mean ratio = 0.70, 90% CI 2-sided [0.55 to 0.88]
Statistical Analysis 18: Comparison: TFV 300mg q.d; Test type: Superiority; p = 0.0046, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum [Note: Comparison of 2nd Trimester vs. Postpartum was not done due to low sample size.]; Geometric mean ratio = 0.80, 90% CI 2-sided [0.72 to 0.89]
Statistical Analysis 19: Comparison: TFV/ATV/RTV Arm 1: 300/300/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum [Note: Comparison of 2nd Trimester vs. Postpartum was not done due to low sample size.]; Geometric mean ratio = 0.66, 90% CI 2-sided [0.52 to 0.85]
Statistical Analysis 20: Comparison: DRV/RTV 800/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 21: Comparison: DRV/RTV 800/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum
Statistical Analysis 22: Comparison: ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d; Test type: Superiority; p > 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 23: Comparison: ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d; Test type: Superiority; p > 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum
Statistical Analysis 24: Comparison: TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 25: Comparison: TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum

5. Primary Outcome: PK Parameter: Area Under the Curve From 0 to 24 Hours (AUC24) With Median (Range) for ARVs and TB Drugs
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. AUC24h (area-under-the-curve from 0 to 24 hours) were determined using the trapezoidal rule.
Time Frame: as for outcome 4
Population: All mothers with intensive pharmacokinetic (PK) results taking the dose under study at that time period (2nd trimester, 3rd trimester or postpartum). Because participants could enter the study at different time period per the study design, they are not expected to have results at every time period. No 2nd trimester data were available for the EFV 600mg q.d. arm.
Measure: Median (Full Range); unit: mg*hour/L
Arm/Group | EFV 600mg q.d. | RPV 25mg q.d.
Number analyzed (Participants) | 25 | 32
mg*hour/L
  2nd Trimester: number analyzed (Participants) | 0 | 18
  2nd Trimester |  | 1.969 [0.867 to 4.987]
  3rd Trimester: number analyzed (Participants) | 25 | 30
  3rd Trimester | 55.4 [13.5 to 220.3] | 1.669 [0.556 to 4.312]
  Postpartum: number analyzed (Participants) | 25 | 28
  Postpartum | 58.3 [22.7 to 214.4] | 2.387 [0.188 to 6.736]
Statistical Analysis 1: Comparison: EFV 600mg q.d; Test type: Superiority; p = 0.07, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.97, 90% CI 2-sided [0.83 to 1.13]
Statistical Analysis 2: Comparison: RPV 25mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.77, 90% CI 2-sided [0.61 to 0.96]
Statistical Analysis 3: Comparison: RPV 25mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.80, 90% CI 2-sided [0.62 to 1.03]

6. Primary Outcome: PK Parameter: Maximum Concentration (Cmax) in mg/L With Median (IQR) for ARVs and TB Drugs
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. Cmax was the maximum observed concentration after a dose.
Time Frame: Measured at 2nd trimester (20-26 wks gestation), 3rd trimester (30-38 wks gestation), and either 2-3 wks, 2-8 wks or 6-12 wks postpartum depending on study arm; Blood samples were drawn pre-dose and at 1, 2, 4, 6, 8,12 (and 24) hours post dosing.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. | DTG 50mg q.d. | DRV/COBI 800/150 mg q.d. | ATV/COBI 300/150 mg q.d. | EFV 600 mg q.d. (Outside THA) | FPV/RTV 700/100mg b.i.d. | ATV/RTV Arm 1: 300/100mg q.d. | TFV 300mg q.d. | TFV/ATV/RTV Arm 1: 300/300/100mg q.d. | EFV 600mg q.d. | DRV/RTV 800/100mg q.d. | DRV/RTV 600/100mg b.i.d. | ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. | TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. | NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d. | IDV/RTV Arm 2: 400/100mg q.d. (Only THA)
Number analyzed (Participants) | 26 | 29 | 29 | 11 | 42 | 29 | 18 | 37 | 20 | 25 | 32 | 34 | 37 | 35 | 18 | 26
mg/L
  2nd Trimester: number analyzed (Participants) | 9 | 15 | 16 | 6 | 15 | 8 | 1 | 4 | 4 | 0 | 15 | 13 | 14 | 17 | 2 | 13
  2nd Trimester | 6.22 [5.30 to 8.42] | 3.62 [2.57 to 4.63] | 4.59 [2.38 to 6.12] | 2.82 [2.65 to 3.65] | 3.87 [2.82 to 5.67] | 5.61 [4.47 to 6.64] | NA [NA to NA] — Only one participant had data for 2nd Trimester. Individual participant level data are not entered due to being potentially identifiable. | 0.250 [0.202 to 0.355] | 1.2 [0.8 to 1.7] |  | 6.77 [4.35 to 7.84] | 5.64 [3.78 to 6.07] | 3.11 [1.95 to 4.06] | 2.73 [1.65 to 4.02] | NA [NA to NA] — Only 2 participants had data available. Data not entered due to extreme small sample size and concerns regarding confidentiality. | 3.89 [3.36 to 4.29]
  3rd Trimester: number analyzed (Participants) | 24 | 28 | 26 | 8 | 42 | 28 | 18 | 37 | 20 | 25 | 30 | 34 | 37 | 32 | 18 | 25
  3rd Trimester | 6.55 [5.38 to 7.43] | 3.54 [2.66 to 4.24] | 3.67 [3.29 to 4.65] | 2.20 [0.94 to 3.35] | 5.13 [3.62 to 5.9] | 5.12 [3.6 to 6.26] | 3.6 [2.8 to 5.1] | 0.245 [0.207 to 0.334] | 2.5 [1.6 to 3] | 5.44 [4.15 to 6.93] | 5.78 [4.31 to 7.29] | 5.53 [4.44 to 7.10] | 4.51 [3.28 to 5.84] | 3.56 [2.28 to 4.32] | 5.1 [4.3 to 6.5] | 3.62 [2.69 to 4.80]
  Postpartum: number analyzed (Participants) | 24 | 22 | 19 | 9 | 40 | 22 | 13 | 32 | 19 | 25 | 23 | 27 | 34 | 34 | 16 | 26
  Postpartum | 8.96 [7.93 to 10.85] | 4.85 [3.83 to 5.97] | 7.04 [5.70 to 10.75] | 3.90 [1.93 to 4.60] | 4.41 [3.38 to 5.79] | 6.75 [4.31 to 9.24] | 4.1 [3 to 5.8] | 0.298 [0.200 to 0.341] | 4.1 [1.7 to 4.5] | 5.10 [3.95 to 5.85] | 8.11 [6.93 to 10.3] | 7.78 [6.11 to 9.54] | 4.52 [2.31 to 5.61] | 5.43 [3.81 to 6.80] | 5.0 [4.2 to 5.9] | 5.37 [4.78 to 7.41]
Statistical Analysis 1: Comparison: DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d; Test type: Superiority; p = 0.148, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.81, 90% CI 2-sided [0.64 to 1.01]
Statistical Analysis 2: Comparison: DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d; Test type: Superiority; p < 0.001, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 0.71, 90% CI 2-sided [0.62 to 0.81]
Statistical Analysis 3: Comparison: DTG 50mg q.d; Test type: Superiority; p = 0.0098, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.74, 90% CI 2-sided [0.61 to 0.89]
Statistical Analysis 4: Comparison: DTG 50mg q.d; Test type: Superiority; p = 0.0025, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 0.75, 90% CI 2-sided [0.64 to 0.88]
Statistical Analysis 5: Comparison: DRV/COBI 800/150 mg q.d; Test type: Superiority; p < 0.0001, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 0.54, 90% CI 2-sided [0.46 to 0.64]
Statistical Analysis 6: Comparison: DRV/COBI 800/150 mg q.d; Test type: Superiority; p = 0.0024, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.56, 90% CI 2-sided [0.41 to 0.76]
Statistical Analysis 7: Comparison: ATV/COBI 300/150 mg q.d; Test type: Superiority; p = 0.438, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.795, 90% CI 2-sided [0.499 to 1.269]
Statistical Analysis 8: Comparison: ATV/COBI 300/150 mg q.d; Test type: Superiority; p = 0.219, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 0.531, 90% CI 2-sided [0.186 to 1.512]
Statistical Analysis 9: Comparison: EFV 600 mg q.d. (Outside THA); Test type: Superiority; p = 0.296, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 1.05, 90% CI 2-sided [0.94 to 1.18]
Statistical Analysis 10: Comparison: EFV 600 mg q.d. (Outside THA); Test type: Superiority; p = 0.007, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 1.26, 90% CI 2-sided [1.01 to 1.56]
Statistical Analysis 11: Comparison: FPV/RTV 700/100mg b.i.d; FPV was analyzed as the form of amprenavir (APV). FPV is the prodrug of APV; Test type: Superiority; p = 0.16, Wilcoxon signed rank test — 2nd Trimester vs Postpartum; Geometric mean of ratio = 0.83, 90% CI 2-sided [0.56 to 1.22]
Statistical Analysis 12: Comparison: FPV/RTV 700/100mg b.i.d; FPV was analyzed in the form of amprenavir (APV). FPV is the prodrug of APV; Test type: Superiority; p = 0.03, Wilcoxson signed rank test; Geometric mean of ratio = 0.74, 90% CI 2-sided [0.58 to 0.93]
Statistical Analysis 13: Comparison: ATV/RTV Arm 1: 300/100mg q.d; This analysis was for ATV; Test type: Superiority; p > 0.05, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum (No comparison was done for 2nd Trimester vs. Postpartum since the sample size for 2nd trimester was 1); Geometric mean of ratio = 0.86, 90% CI 2-sided [0.68 to 1.08]
Statistical Analysis 14: Comparison: TFV 300mg q.d; Test type: Superiority; p = 0.1636, Wilcoxon signed rank test — Third Trimester vs. Postpartum (No comparison was done for Second Trimester vs. Postpartum since only 4 participants had Second Trimester data); Geometric mean of ratio = 0.89, 90% CI 2-sided [0.79 to 1.01]
Statistical Analysis 15: Comparison: TFV/ATV/RTV Arm 1: 300/300/100mg q.d; This analysis was for ATV; Test type: Superiority; p < 0.05, Wilcoxon signed rank test — 3rd Trimester vs Postpartum (No comparison was done for Second Trimester vs. Postpartum since only 4 participants had Second Trimester data); Geometric mean of ratio = 0.69, 90% CI 2-sided [0.53 to 0.91]
Statistical Analysis 16: Comparison: EFV 600mg q.d; Test type: Superiority; p = 0.16, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum (No comparison was done for Second Trimester vs. Postpartum since there was no Second Trimester data available); Geometric mean of ratio = 1.11, 90% CI 2-sided [0.99 to 1.24]
Statistical Analysis 17: Comparison: DRV/RTV 800/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 18: Comparison: DRV/RTV 800/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum
Statistical Analysis 19: Comparison: DRV/RTV 600/100mg b.i.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 20: Comparison: DRV/RTV 600/100mg b.i.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum
Statistical Analysis 21: Comparison: ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d; Test type: Superiority; p > 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 22: Comparison: ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d; Test type: Superiority; p > 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum
Statistical Analysis 23: Comparison: TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 24: Comparison: TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum
Statistical Analysis 25: Comparison: NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d; Test type: Superiority; p = 0.67, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum (No comparison was done for Second Trimester vs. Postpartum since only 2 participants had Second Trimester data); Geometric mean of ratio = 1.06, 90% CI 2-sided [0.85 to 1.34]
Statistical Analysis 26: Comparison: IDV/RTV Arm 2: 400/100mg q.d. (Only THA); Test type: Superiority; p = 0.08, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.73, 90% CI 2-sided [0.59 to 0.91]
Statistical Analysis 27: Comparison: IDV/RTV Arm 2: 400/100mg q.d. (Only THA); Test type: Superiority; p < 0.01, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 0.63, 90% CI 2-sided [0.55 to 0.72]

7. Primary Outcome: PK Parameter: Maximum Concentration (Cmax) in mg/L With Median (Range) for ARVs and TB Drugs
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/L
Arm/Group | LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. | RAL 400mg b.i.d. | ETR 200mg b.i.d. | RPV 25mg q.d.
Number analyzed (Participants) | 33 | 42 | 15 | 32
mg/L
  2nd Trimester: number analyzed (Participants) | 11 | 16 | 5 | 18
  2nd Trimester | 8.4 [7.1 to 10.9] | 2.250 [0.365 to 5.960] | 0.70 [0.44 to 1.05] | 0.145 [0.043 to 0.347]
  3rd Trimester: number analyzed (Participants) | 33 | 41 | 13 | 30
  3rd Trimester | 10.7 [5.8 to 19.1] | 1.770 [0.315 to 7.820] | 1.01 [0.26 to 3.47] | 0.134 [0.049 to 0.267]
  Postpartum: number analyzed (Participants) | 27 | 38 | 8 | 28
  Postpartum | 14.6 [9.8 to 22.8] | 3.035 [0.312 to 12.600] | 0.63 [0.30 to 1.60] | 0.134 [0.048 to 0.407]
Statistical Analysis 1: Comparison: LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d; Test type: Superiority; p < 0.05, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.57, 90% CI 2-sided [0.48 to 0.68]
Statistical Analysis 2: Comparison: LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d; Test type: Superiority; p < 0.05, Wilcoxon signed rank test — 3rd Trimester vs.Postpartum; Geometric mean of ratio = 0.73, 90% CI 2-sided [0.62 to 0.85]
Statistical Analysis 3: Comparison: RAL 400mg b.i.d; Test type: Superiority; p = 0.09, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 4: Comparison: RAL 400mg b.i.d; Test type: Superiority; p = 0.003, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum
Statistical Analysis 5: Comparison: ETR 200mg b.i.d; Test type: Superiority; p = 0.036, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum (No comparison was done for Second Trimester vs. Postpartum since only 5 participants had Second Trimester data); Geometric mean of ratio = 1.34
Statistical Analysis 6: Comparison: RPV 25mg q.d; Test type: Superiority; p > 0.05, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.84, 90% CI 2-sided [0.69 to 1.02]
Statistical Analysis 7: Comparison: RPV 25mg q.d; Test type: Superiority; p > 0.05, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 0.83, 90% CI 2-sided [0.68 to 1.01]

8. Primary Outcome: PK Parameter: Maximum Concentration (Cmax) in ng/mL With Median (IQR) for ARVs and TB Drugs
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | TAF 25mg q.d. | TAF 10mg q.d. w/COBI | TAF 25mg q.d. w/COBI or RTV Boosting | EVG/COBI 150/150mg q.d.
Number analyzed (Participants) | 27 | 31 | 29 | 30
ng/mL
  2nd Trimester: number analyzed (Participants) | 15 | 18 | 12 | 17
  2nd Trimester | 69.7 [50.0 to 112] | 80.4 [57.5 to 121] | 87.8 [44 to 186.5] | 1447.1 [1133.6 to 1579]
  3rd Trimester: number analyzed (Participants) | 27 | 27 | 27 | 26
  3rd Trimester | 96 [63.1 to 112] | 91.2 [51.4 to 136] | 107 [72.9 to 157] | 1432.8 [705.7 to 1570.4]
  Postpartum: number analyzed (Participants) | 25 | 22 | 22 | 25
  Postpartum | 133 [88 to 230] | 98.2 [71.2 to 141] | 141 [51.6 to 244] | 1713.1 [955.7 to 2284.6]
Statistical Analysis 1: Comparison: TAF 25mg q.d; Test type: Superiority; p = 0.14, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.61, 90% CI 2-sided [0.34 to 1.09]
Statistical Analysis 2: Comparison: TAF 25mg q.d; Test type: Superiority; p = 0.002, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 0.64, 90% CI 2-sided [0.50 to 0.81]
Statistical Analysis 3: Comparison: TAF 10mg q.d. w/COBI; Test type: Superiority; p = 0.24, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.77, 90% CI 2-sided [0.49 to 1.23]
Statistical Analysis 4: Comparison: TAF 10mg q.d. w/COBI; Test type: Superiority; p = 0.53, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 0.84, 90% CI 2-sided [0.60 to 1.17]
Statistical Analysis 5: Comparison: TAF 25mg q.d. w/COBI or RTV Boosting; Test type: Superiority; p = 0.2, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.58, 90% CI 2-sided [0.30 to 1.11]
Statistical Analysis 6: Comparison: TAF 25mg q.d. w/COBI or RTV Boosting; Test type: Superiority; p = 0.12, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 0.95, 90% CI 2-sided [0.58 to 1.55]
Statistical Analysis 7: Comparison: EVG/COBI 150/150mg q.d; Test type: Superiority; p = 0.358, Wilcoxon signed rank test — 2nd Trimester vs. Postpartum; Geometric mean of ratio = 0.92, 90% CI 2-sided [0.71 to 1.2]
Statistical Analysis 8: Comparison: EVG/COBI 150/150mg q.d; Test type: Superiority; p = 0.0156, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum; Geometric mean of ratio = 0.72, 90% CI 2-sided [0.55 to 0.93]

9. Primary Outcome: PK Parameter: Maximum Concentration (Cmax) in ng/mL With Median (95% CI) for ARVs and TB Drugs
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: ng/mL
Arm/Group | MVC 150 or 300mg b.i.d.
Number analyzed (Participants) | 18
ng/mL
  2nd Trimester: number analyzed (Participants) | 0
  3rd Trimester: number analyzed (Participants) | 12
  3rd Trimester | 448 [318 to 632]
  Postpartum: number analyzed (Participants) | 10
  Postpartum | 647 [408 to 1025]
Statistical Analysis 1: Comparison: MVC 150 or 300mg b.i.d; Test type: Superiority; p = 0.007, Wilcoxon signed rank test — 3rd Trimester vs. Postpartum (No comparison was done for Second Trimester vs. Postpartum since no Second Trimester data was available); Geometric mean of ratio = 0.7, 90% CI 2-sided [0.58 to 0.85]

10. Primary Outcome: PK Parameter: Trough Concentration (C12) With Median (IQR) for ARVs and TB Drugs
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. Trough concentration was the measured concentration from the 12h post-dose sample after an observed dose.
Time Frame: Measured at 2nd trimester (20-26 wks gestation); 3rd trimester (30-38 gestation); and either 2-3 wks, 2-8 wks, or 6-12 wks postpartum, depending on study arm. Trough concentration was measured 12 hrs after an observed dose.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. | FPV/RTV 700/100mg b.i.d. | DRV/RTV 600/100mg b.i.d. | NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d.
Number analyzed (Participants) | 24 | 29 | 34 | 18
mg/L
  2nd Trimester: number analyzed (Participants) | 9 | 8 | 13 | 18
  2nd Trimester | 2.84 [2.24 to 3.23] | 2.12 [1.39 to 2.67] | 2.12 [1.76 to 2.85] | NA [NA to NA] — PK parameters not calculated for the 2nd trimester
  3rd Trimester: number analyzed (Participants) | 24 | 28 | 34 | 18
  3rd Trimester | 2.52 [2.06 to 2.91] | 1.64 [1.16 to 2.21] | 2.22 [1.68 to 3.26] | 0.47 [0.35 to 1.33]
  Postpartum: number analyzed (Participants) | 24 | 22 | 27 | 16
  Postpartum | 4.51 [3.72 to 5.30] | 2.87 [2.34 to 3.41] | 2.51 [2.04 to 3.27] | 0.52 [0.22 to 0.80]
Statistical Analysis 1: Comparison: DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d; Test type: Superiority; p = 0.109, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.66, 90% CI 2-sided [0.39 to 1.12]
Statistical Analysis 2: Comparison: DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d; Test type: Superiority; p < 0.001, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.58, 90% CI 2-sided [0.49 to 0.69]
Statistical Analysis 3: Comparison: FPV/RTV 700/100mg b.i.d; Test type: Superiority; p = 0.44, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.48, 90% CI 2-sided [0.14 to 1.65]
Statistical Analysis 4: Comparison: FPV/RTV 700/100mg b.i.d; Test type: Superiority; p < 0.001, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.56, 90% CI 2-sided [0.43 to 0.72]
Statistical Analysis 5: Comparison: DRV/RTV 600/100mg b.i.d; Test type: Superiority; p = 0.43, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.83, 90% CI 2-sided [0.63 to 1.10]
Statistical Analysis 6: Comparison: DRV/RTV 600/100mg b.i.d; Test type: Superiority; p = 0.31, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 1.00, 90% CI 2-sided [0.69 to 1.44]
Statistical Analysis 7: Comparison: NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d; Test type: Superiority; p = 0.49, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.90, 90% CI 2-sided [0.71 to 1.16]

11. Primary Outcome: PK Parameter: Trough Concentration (C12) With Median (Range) for ARVs and TB Drugs
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/L
Arm/Group | LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. | RAL 400mg b.i.d. | ETR 200mg b.i.d. | IDV/RTV Arm 2: 400/100mg q.d. (Only THA)
Number analyzed (Participants) | 33 | 42 | 15 | 26
mg/L
  2nd Trimester: number analyzed (Participants) | 11 | 16 | 5 | 13
  2nd Trimester | 3.7 [2.2 to 4.4] | 0.0621 [0.0128 to 0.438] | 0.36 [0.08 to 0.75] | 0.13 [0.07 to 0.23]
  3rd Trimester: number analyzed (Participants) | 33 | 41 | 13 | 25
  3rd Trimester | 5.1 [1.5 to 12.2] | 0.064 [0.0114 to 0.607] | 0.48 [0.08 to 1.94] | 0.13 [0.07 to 0.60]
  Postpartum: number analyzed (Participants) | 27 | 38 | 8 | 26
  Postpartum | 7.2 [2.8 to 21] | 0.0797 [0.0199 to 1.340] | 0.38 [0.07 to 1.14] | 0.28 [0.14 to 0.71]
Statistical Analysis 1: Comparison: LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.45, 90% CI 2-sided [0.32 to 0.63]
Statistical Analysis 2: Comparison: LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.72, 90% CI 2-sided [0.58 to 0.88]
Statistical Analysis 3: Comparison: RAL 400mg b.i.d; Test type: Superiority; p = 0.02, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.42, 90% CI 2-sided [0.23 to 0.78]
Statistical Analysis 4: Comparison: RAL 400mg b.i.d; Test type: Superiority; p = 0.3, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.78, 90% CI 2-sided [0.56 to 1.08]
Statistical Analysis 5: Comparison: ETR 200mg b.i.d; Test type: Superiority; p = 0.036, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum [Note: Comparison of 2nd Trimester vs. Postpartum was not done due to low sample size.]; Geometric mean ratio = 1.41
Statistical Analysis 6: Comparison: IDV/RTV Arm 2: 400/100mg q.d. (Only THA); Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.41, 90% CI 2-sided [0.32 to 0.52]
Statistical Analysis 7: Comparison: IDV/RTV Arm 2: 400/100mg q.d. (Only THA); Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.48, 90% CI 2-sided [0.41 to 0.57]

12. Primary Outcome: PK Parameter: Trough Concentration (C12) With Geometric Mean (95% CI) for ARVs and TB Drugs
Description: as for outcome 10
Time Frame: Measured at 2nd trimester (20-26 wks gestation), 3rd trimester (30-38 wks gestation), and either 2-3 wks, 2-8 wks or 6-12 wks postpartum depending on study arm. Trough concentration was measured 12 hrs after an observed dose.
Population: All mothers with intensive pharmacokinetic (PK) results taking the dose under study at that time period (2nd trimester, 3rd trimester or postpartum). Because participants could enter the study at different time period per the study design, they are not expected to have results at every time period. No 2nd trimester data were available for the MVC 150 or 300mg b.i.d. arm.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | MVC 150 or 300mg b.i.d.
Number analyzed (Participants) | 18
ng/mL
  2nd Trimester: number analyzed (Participants) | 0
  3rd Trimester: number analyzed (Participants) | 12
  3rd Trimester | 108 [81 to 145]
  Postpartum: number analyzed (Participants) | 10
  Postpartum | 128 [89 to 184]
Statistical Analysis 1: Comparison: MVC 150 or 300mg b.i.d; Test type: Superiority; p = 0.10, t-test, 2 sided — 3rd Trimester vs. Postpartum; Paired sample t-test on natural log-transformed PK parameter; Geometric mean ratio = 0.85, 90% CI 2-sided [0.72 to 1.01]

13. Primary Outcome: PK Parameter: Trough Concentration (C24) With Median (IQR) for ARVs and TB Drugs
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. Trough concentration was the measured concentration from the 24h post-dose sample after an observed dose.
  For the TAF 25 mg q.d., 10 mg q.d. w/COBI, and 25 mg q.d. w/COBI or RTV boosting arms, samples were all below the limit of quantification and statistical analyses were not conducted.
Time Frame: Measured at 2nd trimester (20-26 wks gestation), 3rd trimester (30-38 wks gestation), and either 2-3 wks, 2-8 wks or 6-12 wks postpartum depending on study arm. Trough concentration was measured 24 hrs after an observed dose.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | DTG 50mg q.d. | TAF 25mg q.d. | TAF 10mg q.d. w/COBI | TAF 25mg q.d. w/COBI or RTV Boosting | EVG/COBI 150/150mg q.d. | DRV/COBI 800/150 mg q.d. | ATV/COBI 300/150 mg q.d. | EFV 600 mg q.d. (Outside THA) | ATV/RTV Arm 1: 300/100mg q.d. | TFV 300mg q.d. | TFV/ATV/RTV Arm 1: 300/300/100mg q.d. | DRV/RTV 800/100mg q.d. | ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. | TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d.
Number analyzed (Participants) | 29 | 27 | 31 | 29 | 30 | 29 | 11 | 42 | 18 | 37 | 20 | 32 | 37 | 35
mg/L
  2nd Trimester: number analyzed (Participants) | 15 | 15 | 18 | 12 | 17 | 16 | 6 | 15 | 1 | 4 | 4 | 15 | 14 | 17
  2nd Trimester | 0.73 [0.63 to 1.34] | 0.00195 [0.00195 to 0.00195] | 0.00195 [0.00195 to 0.00195] | 0.00195 [0.00195 to 0.00195] | 0.0258 [0.0179 to 0.0672] | 0.33 [0.045 to 0.47] | 0.21 [0.16 to 0.28] | 1.49 [1.14 to 2.23] | 2.0 [NA to NA] — IQR could not be estimated since only one Ctrough was calculated | 0.039 [0.034 to 0.049] | 0.3 [0.2 to 0.4] | 0.99 [0.43 to 1.81] | 0.49 [0.26 to 0.78] | 0.44 [0.28 to 0.59]
  3rd Trimester: number analyzed (Participants) | 28 | 27 | 26 | 27 | 26 | 26 | 8 | 42 | 18 | 37 | 20 | 30 | 37 | 32
  3rd Trimester | 0.93 [0.68 to 1.34] | 0.00195 [0.00195 to 0.00195] | 0.00195 [0.00195 to 0.00195] | 0.00195 [0.00195 to 0.00195] | 0.0487 [0.0140 to 0.0751] | 0.27 [0.045 to 0.63] | 0.21 [0.11 to 0.56] | 1.48 [1.10 to 2.61] | 0.7 [0.5 to 1.1] | 0.054 [0.040 to 0.070] | 0.5 [0.4 to 0.7] | 1.17 [0.73 to 1.72] | 0.71 [0.47 to 1.0] | 0.57 [0.39 to 0.81]
  Postpartum: number analyzed (Participants) | 22 | 26 | 23 | 22 | 25 | 19 | 9 | 40 | 13 | 32 | 19 | 23 | 34 | 34
  Postpartum | 1.28 [0.80 to 1.95] | 0.00195 [0.00195 to 0.00195] | 0.00195 [0.00195 to 0.00195] | 0.00195 [0.00195 to 0.00195] | 0.3771 [0.2285 to 0.5688] | 1.43 [0.73 to 1.86] | 0.61 [0.42 to 1.03] | 1.94 [1.28 to 3.09] | 1.2 [1.1 to 2.0] | 0.061 [0.045 to 0.079] | 0.8 [0.6 to 1.2] | 2.78 [2.05 to 2.98] | 0.90 [0.39 to 1.33] | 1.26 [0.69 to 1.95]
Statistical Analysis 1: Comparison: DTG 50mg q.d; Test type: Superiority; p = 0.0039, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.49, 90% CI 2-sided [0.35 to 0.68]
Statistical Analysis 2: Comparison: DTG 50mg q.d; Test type: Superiority; p = 0.0062, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.66, 90% CI 2-sided [0.52 to 0.84]
Statistical Analysis 3: Comparison: EVG/COBI 150/150mg q.d; Test type: Superiority; p < 0.10, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 4: Comparison: EVG/COBI 150/150mg q.d; Test type: Superiority; p < 0.10, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum
Statistical Analysis 5: Comparison: DRV/COBI 800/150 mg q.d; Test type: Superiority; p < 0.10, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.15, 90% CI 2-sided [0.08 to 0.30]
Statistical Analysis 6: Comparison: DRV/COBI 800/150 mg q.d; Test type: Superiority; p < 0.10, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.21, 90% CI 2-sided [0.12 to 0.36]
Statistical Analysis 7: Comparison: ATV/COBI 300/150 mg q.d; Test type: Superiority; p < 0.10, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.32, 90% CI 2-sided [0.20 to 0.51]
Statistical Analysis 8: Comparison: ATV/COBI 300/150 mg q.d; Test type: Superiority; p > 0.10, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.32, 90% CI 2-sided [0.11 to 0.94]
Statistical Analysis 9: Comparison: EFV 600 mg q.d. (Outside THA); Test type: Other; p = 0.079, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.87, 90% CI 2-sided [0.78 to 0.97]
Statistical Analysis 10: Comparison: EFV 600 mg q.d. (Outside THA); Test type: Superiority; p = 0.01, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.92, 90% CI 2-sided [0.77 to 1.09]
Statistical Analysis 11: Comparison: ATV/RTV Arm 1: 300/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum [Note: Comparison of 2nd Trimester vs. Postpartum was not done due to low sample size.]; Geometric mean ratio = 0.51, 90% CI 2-sided [0.37 to 0.72]
Statistical Analysis 12: Comparison: TFV 300mg q.d; Test type: Superiority; p = 0.0325, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum [Note: Comparison of 2nd Trimester vs. Postpartum was not done due to low sample size.]; Geometric mean ratio = 0.82, 90% CI 2-sided [0.71 to 0.96]
Statistical Analysis 13: Comparison: TFV/ATV/RTV Arm 1: 300/300/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum [Note: Comparison of 2nd Trimester vs. Postpartum was not done due to low sample size.]; Geometric mean ratio = 0.65, 90% CI 2-sided [0.54 to 0.77]
Statistical Analysis 14: Comparison: DRV/RTV 800/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 15: Comparison: DRV/RTV 800/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum
Statistical Analysis 16: Comparison: ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d; Test type: Superiority; p > 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 17: Comparison: ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d; Test type: Superiority; p > 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum
Statistical Analysis 18: Comparison: TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum
Statistical Analysis 19: Comparison: TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum

14. Primary Outcome: PK Parameter: Trough Concentration (C24) With Median (Range) for ARVs and TB Drugs
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. Trough concentration was the measured concentration from the 24h post-dose sample after an observed dose.
Time Frame: as for outcome 13
Population: as for outcome 5
Measure: Median (Full Range); unit: mg/L
Arm/Group | EFV 600mg q.d. | RPV 25mg q.d.
Number analyzed (Participants) | 25 | 32
mg/L
  2nd Trimester: number analyzed (Participants) | 0 | 18
  2nd Trimester |  | 0.063 [0.037 to 0.225]
  3rd Trimester: number analyzed (Participants) | 25 | 30
  3rd Trimester | 1.60 [0.23 to 8.13] | 0.056 [0.010 to 0.181]
  Postpartum: number analyzed (Participants) | 25 | 28
  Postpartum | 2.05 [0.31 to 8.43] | 0.081 [0.010 to 0.299]
Statistical Analysis 1: Comparison: EFV 600mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.88, 90% CI 2-sided [0.73 to 1.06]
Statistical Analysis 2: Comparison: RPV 25mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 2nd Trimester vs. Postpartum; Geometric mean ratio = 0.70, 90% CI 2-sided [0.55 to 0.90]
Statistical Analysis 3: Comparison: RPV 25mg q.d; Test type: Superiority; p < 0.05, Wilcoxon signed-rank test — 3rd Trimester vs. Postpartum; Geometric mean ratio = 0.84, 90% CI 2-sided [0.57 to 1.23]

15. Primary Outcome: Number of Women Who Met PK Target of Area Under the Curve (AUC) for ARVs
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. AUC (area under the curve) were determined using the linear trapezoidal rule. See PK target in the Protocol Appendix V.
Time Frame: Measured at 2nd trimester (20-26 wks gestation), 3rd trimester (30-38 wks gestation), and either 2-3 wks, 2-8 wks or 6-12 wks postpartum depending on study arm. Blood samples were drawn pre-dose and at 1, 2, 4, 6, 8, 12 (and 24) hours post dosing.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. | DTG 50mg q.d. | TAF 25mg q.d. | TAF 10mg q.d. w/COBI | TAF 25mg q.d. w/COBI or RTV Boosting | EVG/COBI 150/150mg q.d. | DRV/COBI 800/150 mg q.d. | ATV/COBI 300/150 mg q.d. | EFV 600 mg q.d. (Outside THA) | FPV/RTV 700/100mg b.i.d. | ATV/RTV Arm 1: 300/100mg q.d. | TFV 300mg q.d. | TFV/ATV/RTV Arm 1: 300/300/100mg q.d. | EFV 600mg q.d. | LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. | RAL 400mg b.i.d. | ETR 200mg b.i.d. | MVC 150 or 300mg b.i.d. | DRV/RTV 800/100mg q.d. | DRV/RTV 600/100mg b.i.d. | ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. | TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. | NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d. | IDV/RTV Arm 2: 400/100mg q.d. (Only THA) | RPV 25mg q.d.
Number analyzed (Participants) | 26 | 29 | 27 | 31 | 29 | 30 | 29 | 11 | 42 | 29 | 18 | 37 | 20 | 25 | 33 | 42 | 15 | 18 | 32 | 34 | 37 | 35 | 18 | 26 | 32
Participants
  2nd Trimester: number analyzed (Participants) | 8 | 15 | 15 | 18 | 12 | 17 | 16 | 6 | 15 | 8 | 1 | 4 | 4 | 0 | 11 | 16 | 5 | 0 | 15 | 13 | 14 | 17 | 2 | 13 | 15
  2nd Trimester | 7 | 9 | 13 | 15 | 10 | 8 | 3 | 1 | 12 | 8 | 1 | 2 | 1 |  | 9 | 11 | 5 |  | 9 | 7 | 8 | 7 | NA — Only 2 participants had data available. Data not entered due to extreme small sample size and concerns regarding confidentiality. | 10 | 14
  3rd Trimester: number analyzed (Participants) | 23 | 28 | 27 | 27 | 27 | 26 | 26 | 9 | 41 | 28 | 18 | 37 | 20 | 25 | 33 | 41 | 13 | 11 | 30 | 34 | 37 | 32 | 18 | 25 | 28
  3rd Trimester | 16 | 20 | 23 | 23 | 24 | 10 | 4 | 2 | 33 | 26 | 12 | 27 | 11 | 20 | 30 | 33 | 13 | 8 | 19 | 19 | 29 | 23 | 15 | 19 | 26
  Postpartum: number analyzed (Participants) | 23 | 23 | 25 | 24 | 22 | 25 | 20 | 9 | 40 | 22 | 13 | 32 | 19 | 25 | 27 | 38 | 8 | 8 | 24 | 27 | 34 | 34 | 16 | 26 | 28
  Postpartum | 22 | 23 | 24 | 22 | 18 | 18 | 14 | 5 | 34 | 22 | 12 | 27 | 12 | 21 | 27 | 30 | 7 | 7 | 22 | 22 | 27 | 32 | 14 | 26 | 25

16. Primary Outcome: Number of Women Who Met PK Target of Maximum Concentration (Cmax) for First Line TB Drugs
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. Cmax was the maximum observed concentration after a dose. See PK target in Protocol Appendix V.
  The reporting groups for this outcome reflect the drug being analyzed and are therefore not mutually exclusive.
  No results are available for LPV/RTV 800/200mg b.i.d. and at least one 1st line TB drug arm due to extremely low enrollment.
Time Frame: as for outcome 15
Population: All mothers with intensive pharmacokinetic (PK) results taking the dose under study at that time period (2nd trimester, 3rd trimester or postpartum). Because participants could enter the study at different time period per the study design, they are not expected to have results at every time period. No data are available for LPV/RTV 800/200mg b.i.d. and at least one 1st line TB drug due to extremely low enrollment.
Measure: Count of Participants; unit: Participants
Groups:
- EFV 600mg q.d. and at Least One 1st Line TB Drug - Isoniazid: HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz (EFV) 600mg q.d.and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  This group is for the participants who received isoniazid.
- EFV 600mg q.d. and at Least One 1st Line TB Drug - Rifampicin: HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz (EFV) 600mg q.d.and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w
  This group is for the participants who received rifampicin.
- EFV 600mg q.d. and at Least One 1st Line TB Drug - Pyrazinamide: HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz (EFV) 600mg q.d.and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  This group is for the participants who received pyrazinamide.
- EFV 600mg q.d. and at Least One 1st Line TB Drug - Ethambutol: HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz (EFV) 600mg q.d.and
  TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  This group is for the participants who received ethambutol.
- No ARVs and at Least Two 1st Line TB Drugs - Isoniazid: HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following first line TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  This group is for the participants who recieved isoniazid.
- No ARVs and at Least Two 1st Line TB Drugs - Rifampicin: HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following first line TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  This group is for the participants who recieved rifampicin.
- No ARVs and at Least Two 1st Line TB Drugs - Pyrazinamide: HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following first line TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
  This group is for the participants who received pyrazinamide.
- No ARVs and at Least Two 1st Line TB Drugs - Ethambutol: HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following first line TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w
  This group is for the participants who received ethambutol.
Arm/Group | LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug | EFV 600mg q.d. and at Least One 1st Line TB Drug - Isoniazid | EFV 600mg q.d. and at Least One 1st Line TB Drug - Rifampicin | EFV 600mg q.d. and at Least One 1st Line TB Drug - Pyrazinamide | EFV 600mg q.d. and at Least One 1st Line TB Drug - Ethambutol | No ARVs and at Least Two 1st Line TB Drugs - Isoniazid | No ARVs and at Least Two 1st Line TB Drugs - Rifampicin | No ARVs and at Least Two 1st Line TB Drugs - Pyrazinamide | No ARVs and at Least Two 1st Line TB Drugs - Ethambutol
Number analyzed (Participants) | 0 | 22 | 22 | 8 | 8 | 24 | 26 | 13 | 16
Participants
  2nd Trimester: number analyzed (Participants) | 0 | 12 | 12 | 4 | 4 | 14 | 16 | 6 | 8
  2nd Trimester |  | 5 | 4 | 4 | 3 | 11 | 8 | 6 | 4
  3rd Trimester: number analyzed (Participants) | 0 | 20 | 20 | 4 | 5 | 19 | 20 | 9 | 11
  3rd Trimester |  | 16 | 6 | 4 | 2 | 13 | 8 | 9 | 8
  Postpartum: number analyzed (Participants) | 0 | 13 | 13 | 1 | 1 | 12 | 13 | 2 | 4
  Postpartum |  | 7 | 6 | 1 | 0 | 9 | 6 | 2 | 4

17. Primary Outcome: Plasma Concentration for Contraceptives
Description: Serum concentrations of the contraceptives. Note that no historical controls were provided by team pharmacologists and thus no comparisons were done for contraceptive concentrations in women using hormonal contraceptives and selected ARV drugs as compared to historical controls not using those ARV drugs.
Time Frame: Measured at 6-7 weeks after contraceptive initiation postpartum
Population: HIV-infected women 2-12 weeks (14-84 days) post-delivery receiving ARV drug combinations AND starting postpartum contraceptives as listed in the protocol with intensive PK results.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | ATV/RTV/TFV 300/100/300mg q.d. With ENG | LPV/RTV 400/100 b.i.d. With ENG | EFV 600mg q.d. With ENG
Number analyzed (Participants) | 22 | 26 | 26
pg/mL | 604 [436 to 838] | 428 [340 to 563] | 125 [41.5 to 202]

18. Primary Outcome: Area Under the Curve From 0 to 12 Hours (AUC12) of ARVs for Contraceptive Arms
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. AUC12h (area-under-the-curve from 0 to 12 hours) were determined using the linear trapezoidal rule.
Time Frame: Measured at 2-12 wks postpartum before contraceptive initiation and 6-7 wks after contraceptive initiation. Blood samples were drawn pre-dose and at 0, 1, 2, 6, 8 and 12 hours post dosing.
Population: as for outcome 17
Measure: Median (Full Range); unit: mcg*hr/mL
Arm/Group | LPV/RTV 400/100 b.i.d. With ENG
Number analyzed (Participants) | 26
mcg*hr/mL
  Before contraceptive initiation | 115.97 [15.78 to 259.48]
  After contraceptive initiation | 100.20 [3.39 to 159.93]
Statistical Analysis 1: Comparison: LPV/RTV 400/100 b.i.d. With ENG; The statistical analysis is for LPV PK; Test type: Superiority; p = 0.114, Wilcoxon signed rank test — Before ENG initiation vs. after ENG initiation; Geometric mean of ratio = 1.24, 90% CI 2-sided [0.97 to 1.59]

19. Primary Outcome: Area Under the Curve From 0 to 24 Hours (AUC24) of ARVs for Contraceptive Arms
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods. AUC24h (area-under-the-curve from 0 to 24 hours) were determined using the linear trapezoidal rule.
Time Frame: Measured at 2-12 wks postpartum before contraceptive initiation and 6-7 wks after contraceptive initiation. Blood samples were drawn pre-dose and at 0, 1, 2, 6, 8, 12, and 24 hours post dosing.
Population: HIV-infected women 2-12 weeks (14-84 days) post-delivery receiving one of the ARV drug combinations AND starting postpartum contraceptives as listed in the protocol with intensive PK results.
Measure: Median (Full Range); unit: mcg*hr/mL
Arm/Group | ATV/RTV/TFV 300/100/300mg q.d. With ENG | EFV 600mg q.d. With ENG
Number analyzed (Participants) | 22 | 26
mcg*hr/mL
  Before contraceptive initiation | 53.96 [8.74 to 157.30] | 53.64 [26.29 to 216.55]
  After contraceptive initiation | 55.25 [9.47 to 157.57] | 56.65 [26.28 to 299.55]
Statistical Analysis 1: Comparison: ATV/RTV/TFV 300/100/300mg q.d. With ENG; The statistical test is for ATV PK; Test type: Superiority; p = 0.367, Wilcoxon signed rank test — Before ENG initiation vs. after ENG initiation; Geometric mean of ratio = 1.10, 90% CI 2-sided [0.84 to 1.44]
Statistical Analysis 2: Comparison: EFV 600mg q.d. With ENG; The statistical test is for EFV PK; Test type: Superiority; p = 0.561, Wilcoxon signed rank test; Before ENG initiation vs. after ENG initiation; Geometric mean of ratio = 1.02, 90% CI 2-sided [0.92 to 1.13]

20. Secondary Outcome: PK Parameter: Cord/Maternal Blood Concentration Ratio With Median (IQR) for ARVs and TB Drugs
Description: Cord blood and maternal plasma concentrations were collected and measured at delivery, and compared as a ratio.
Time Frame: Measured at time of delivery with single cord blood and single maternal plasma sample.
Population: All participants with cord blood drawn immediately after the cord was clamped and maternal blood samples drawn at the time the cord was clamped at delivery.
Measure: Median (Inter-Quartile Range); unit: unitless
Arm/Group | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. | DTG 50mg q.d. | EVG/COBI 150/150mg q.d. | DRV/COBI 800/150 mg q.d. | ATV/COBI 300/150 mg q.d. | TFV 300mg q.d.
Number analyzed (Participants) | 16 | 18 | 12 | 13 | 6 | 28
unitless | 0.15 [0.12 to 0.17] | 1.25 [1.07 to 1.40] | 0.91 [0.65 to 1.03] | 0.07 [0.03 to 0.15] | 0.07 [0.02 to 0.19] | 0.88 [0.76 to 1.03]

21. Secondary Outcome: PK Parameter: Cord/Maternal Blood Concentration Ratio With Median (Range) for ARVs and TB Drugs
Description: Cord blood and maternal plasma concentrations were collected and measured at delivery, and compared as a ratio. For arms with zero overall participants analyzed, samples were below the limit of quantification and ratios could not be calculated.
Time Frame: Measured at time of delivery with single cord blood and single maternal plasma sample.
Population: All participants with cord blood drawn immediately after the cord was clamped and maternal blood samples drawn at the time the cord was clamped at delivery.
  Notes: a) Ratios were not calculated for the TAF 25mg q.d. and TAF 25mg q.d. w/COBI or RTV Boosting arms since all cord blood samples were below the lower limit of quantification. b)These arms were combined for analysis: (1) ATV/RTV 300/100mg q.d. & TFV/ATV/RTV 300/300/100mg q.d. and (2) DRV/RTV 800/100mg q.d. & DRV/RTV 600/100mg b.i.d.
Measure: Median (Full Range); unit: unitless
Groups:
- ATV/RTV 300/100mg q.d. or TFV/ATV/RTV 300/300/100mg q.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received atazanavir/ritonavir (ATV/RTV) 300/100 mg once a day or tenofovir/atazanavir/ritonavir (TFV/ATV/RTV) 300/300/100 mg once a day atazanavir/ritonavir dosage #1: atazanavir/ritonavir 300/100 mg once a day atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
- DRV/RTV 800/100mg q.d. or DRV/RTV 600/100mg b.i.d.: HIV-infected pregnant women ≥ 20 weeks gestation who received darunavir/ritonavir (DRV/RTV) 800/100 mg once a day or darunavir/ritonavir (DRV/RTV) 600/100 mg twice a day
  darunavir/ritonavir dosage #1: darunavir/ritonavir twice daily 600/100 mg b.i.d.
  darunavir/ritonavir dosage #4: darunavir/ritonavir once daily 800/100 mg q.d.
Arm/Group | TAF 10mg q.d. w/COBI | EFV 600 mg q.d. (Outside THA) | EFV 600mg q.d. | LPV/RTV Arm 3: 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. | RAL 400mg b.i.d. | ETR 200mg b.i.d. | MVC 150 or 300mg b.i.d. | ATV/RTV Arm 2: 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. | TFV/ATV/RTV Arm 2: 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. | NFV Arm 2: 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d. | IDV/RTV Arm 2: 400/100mg q.d. (Only THA) | RPV 25mg q.d. | ATV/RTV 300/100mg q.d. or TFV/ATV/RTV 300/300/100mg q.d. | DRV/RTV 800/100mg q.d. or DRV/RTV 600/100mg b.i.d.
Number analyzed (Participants) | 1 | 17 | 23 | 26 | 29 | 6 | 10 | 27 | 28 | 10 | 19 | 19 | 29 | 28
unitless | 0.97 [NA to NA] — Range not estimated since only one ratio was calculated | 0.67 [0.36 to 0.95] | 0.49 [0.37 to 0.74] | 0.2 [0.04 to 0.97] | 1.5 [0.1 to 4.7] | 0.52 [0.19 to 4.25] | 0.33 [0.03 to 0.56] | 0.14 [0.05 to 0.84] | 0.16 [0.03 to 4.08] | 0.19 [0.16 to 0.92] | 0.12 [0.05 to 0.23] | 0.55 [0.3 to 0.8] | 0.18 [0.04 to 0.45] | 0.18 [0 to 0.82]

22. Secondary Outcome: Pharmacokinetic (PK) Parameter: Infant Plasma Washout Half-life (T1/2) of ARVs and TB Drugs
Description: Infant plasma concentrations were collected and measured during the first 9 days of life. Half-life is defined as 0.693/k, where k, the elimination rate constant, is the slope of the decline in concentrations.
Time Frame: Infant plasma samples at 2-10, 18-28, 36-72 hours and 5-9 days after birth.
Population: All infants who met the requirement for washout PK sampling (as specified in Protocol Section 4.4) with plasma samples drawn after delivery.
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | DTG 50mg q.d. | EVG/COBI 150/150mg q.d. | DRV/COBI 800/150 mg q.d. | EFV 600 mg q.d. (Outside THA)
Number analyzed (Participants) | 16 | 17 | 26 | 18
hour | 32.8 [25.9 to 35.9] | 7.6 [6.3 to 10.2] | NA [NA to NA] — Due to low placental transfer, infant washout elimination could not be assessed. | 65.6 [40.6 to 128.7]

23. Secondary Outcome: Pharmacokinetic (PK) Parameter: Infant Plasma Washout Concentration of ARVs and TB Drugs
Description: Infant plasma concentrations were collected and measured during the first 9 days of life.
Time Frame: Blood samples were collected at 2-10, 18-28, 36-72 hours and 5-9 days after birth.
Population: All infants who met the requirements for washout PK sampling (as specified in Protocol Section 4.4) with plasma samples drawn after delivery. Infants don't need to contribute to all time points to be included. For DRV/COBI 800/150mg q.d. arm, infants with concentrations below detection limit were not summarized.
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | DTG 50mg q.d. | EVG/COBI 150/150mg q.d. | DRV/COBI 800/150 mg q.d. | EFV 600 mg q.d. (Outside THA)
Number analyzed (Participants) | 22 | 27 | 26 | 23
mcg/mL
  2-10 hours after birth: number analyzed (Participants) | 17 | 24 | 6 | 18
  2-10 hours after birth | 1.73 [1.33 to 2.41] | 0.132 [0.024 to 0.396] | 0.35 [0.24 to 2.09] | 1.1 [0.8 to 1.5]
  18-28 hours after birth: number analyzed (Participants) | 18 | 25 | 4 | 21
  18-28 hours after birth | 1.53 [1.04 to 1.91] | 0.032 [0.012 to 0.088] | 1.43 [1.34 to 1.58] | 1.0 [0.8 to 1.2]
  36-72 hours after birth: number analyzed (Participants) | 17 | 24 | 4 | 20
  36-72 hours after birth | 1.00 [0.66 to 1.65] | 0.005 [0.005 to 0.011] | 1.87 [0.92 to 2.20] | 0.9 [0.6 to 1.4]
  5-9 days after birth: number analyzed (Participants) | 17 | 23 | 4 | 22
  5-9 days after birth | 0.06 [0.04 to 0.14] | 0.005 [0.005 to 0.005] | 1.72 [0.99 to 2.54] | 0.4 [0.2 to 0.9]

24. Other Pre Specified Outcome: ARV Concentrations in Plasma
Description: The original study protocol listed this PK parameter under primary outcome measures. However, this PK parameter was intended for potential supporting analyses and thus belong with Other outcome measures (see SAP).
Time Frame: Measured at intensive PK visit
Reporting Status: Not Posted

25. Other Pre Specified Outcome: ARV Concentrations in Vaginal Secretions
Description: The original study protocol listed this PK parameter under secondary outcome measures. However, this PK parameter was intended for potential supporting analyses and thus belongs with Other outcome measures (see SAP).
Time Frame: Measured at intensive PK visit
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Drug Parameter: Half-life (t1/2)
Description: The original study protocol listed this PK parameter under primary outcome measures. However, this PK parameter was intended for potential supporting analyses and thus belongs with Other outcome measures (see SAP).
Time Frame: Measured at intensive PK visit. Timing of intensive PK visit depends on participant's study arm; may occur during 2nd trimester (20-26 wks gestation); 3rd trimester (30-38 wks gestation); and either 2-3 wks, 2-8 wks, or 6-12 wks postpartum.
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Drug Parameter: Volume of Distribution Over Systemic Availability (V/F)
Description: as for outcome 26
Time Frame: Measured at intensive PK visit. Timing of intensive PK visit depends on participant's study arm; may occur during 2nd trimester (20-26 wks gestation); 3rd trimester (30-38 wks gestation); and either 2-3 weeks, 2-8 wks, or 6-12 wks postpartum.
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Drug Parameter: Clearance Over Systemic Availability (Cl/F)
Description: as for outcome 26
Time Frame: as for outcome 26
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Drug Parameter: Time After Administration of Drug When Maximum Plasma Concentration is Reached (Tmax)
Description: as for outcome 26
Time Frame: as for outcome 26
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Drug Parameter: Minimum Concentration (Cmin)
Description: as for outcome 26
Time Frame: as for outcome 27
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Drug Parameter: Pre-dose Concentration (Cdose)
Description: as for outcome 26
Time Frame: as for outcome 26
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Adverse Events of Grade 3 or Higher
Description: The original study protocol listed all non-primary outcome measures under secondary outcome measures without distinguishing between secondary vs other outcome measures. This outcome measure was intended for potential supporting analyses which were not conducted (see SAP).
  See Adverse events section for adverse events.
Time Frame: Measured through 24 weeks postpartum
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Infant Neurological Events of Grade 1 or Higher
Description: as for outcome 32
Time Frame: Measured through 24 weeks of life
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Adverse Pregnancy Outcome: Preterm Birth
Description: as for outcome 32
Time Frame: Measured through delivery
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Adverse Pregnancy Outcome: Low Birth Weight
Description: as for outcome 32
Time Frame: Measured at delivery
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Adverse Pregnancy Outcome: Fetal Demise
Description: as for outcome 32
Time Frame: Measured through 24 weeks postpartum
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Adverse Pregnancy Outcome: Congenital Anomalies
Description: The original study protocol listed all non-primary outcome measures under secondary outcome measures without distinguishing between secondary vs other outcome measures. This outcome measure was intended for potential supporting analyses which werenot conducted (see SAP).
  See Adverse events section for adverse events.
Time Frame: Measured through 24 weeks of life
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Infant HIV Infection Status
Description: The original study protocol listed all non-primary outcome measures under secondary outcome measures without distinguishing between secondary vs other outcome measures. This outcome measure was intended for potential supporting analyses which were not conducted (see SAP).
Time Frame: Measured through 24 weeks of life
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Ratio of Unbound/Total Drug Concentrations
Description: as for outcome 38
Time Frame: Measured at time of delivery
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Rate of Detection of Study Drugs in Vaginal Secretions
Description: as for outcome 38
Time Frame: Measured at intensive PK visit
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Ratio of Vaginal Drug Concentrations to Simultaneous Blood Concentrations
Description: as for outcome 38
Time Frame: Measured at intensive PK visit
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Rate of Detection of HIV RNA/DNA in Vaginal Secretions and Comparison to Level in Blood
Description: as for outcome 38
Time Frame: Measured at intensive PK visit
Reporting Status: Not Posted

43. Other Pre Specified Outcome: ARV Exposure (as Measured by Area Under the Curve or Other PK Parameters) During Pregnancy and Postpartum According to Genotype
Description: as for outcome 38
Time Frame: Measured at intensive PK visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From study entry to the end of study follow-up: • HIV-infected pregnant women without TB: entry to 6-2 weeks after delivery with the exception of women on DRV/r who will be from entry to 2-3 weeks after delivery; • Women receiving TB treatment: entry to 2-8 weeks after delivery; • Postpartum women: entry to 6-7 weeks after the initiation of hormonal contraceptives; • Infants: birth to16-24 weeks of life.
Description: All adverse events including diagnoses, labs and signs/symptoms after study entry for mothers; all diagnoses, labs and signs/symptoms after birth for infants (AEs were summarized separately for moms and infants). The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, dated July 2017 was followed.
Groups:
- ABC 300mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received abacavir 300mg twice a day abacavir: abacavir 300mg twice a day
- ATV/COBI 300/150 mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received atazanavir/cobicistat 300/150 mg q.d.
  atazanavir/cobicistat: atazanavir/cobicistat 300/150 mg q.d.
- ATV/COBI 300/150 mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received atazanavir/cobicistat 300/150 mg q.d.
  atazanavir/cobicistat: atazanavir/cobicistat 300/150 mg q.d.
- ATV/RTV 300/100mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received atazanavir/ritonavir 300/100 mg once a day atazanavir/ritonavir dosage #1: atazanavir/ritonavir 300/100 mg once a day
- ATV/RTV 300/100mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received atazanavir/ritonavir 300/100 mg once a day atazanavir/ritonavir dosage #1: atazanavir/ritonavir 300/100 mg once a day
- ATV/RTV 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received atazanavir/ritonavir 300/100 mg once a day until 30 weeks gestation then 400/100 mg once a day until postpartum hospital discharge; then 300/100 mg once a day after postpartum hospital discharge until 2 week postpartum PK samples drawn atazanavir/ritonavir dosage #1: atazanavir/ritonavir 300/100 mg once a day atazanavir/ritonavir dosage #2: atazanavir/ritonavir 400/100mg once a day
- ATV/RTV 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received atazanavir/ritonavir 300/100 mg once a day until 30 weeks gestation then 400/100 mg once a day until postpartum hospital discharge; then 300/100 mg once a day after postpartum hospital discharge until 2 week postpartum PK samples drawn atazanavir/ritonavir dosage #1: atazanavir/ritonavir 300/100 mg once a day atazanavir/ritonavir dosage #2: atazanavir/ritonavir 400/100mg once a day
- ATV/RTV/TFV 300/100/300mg q.d. With 30-35ug EE MOTHER: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received atazanavir/ritonavir/tenofovir 300/100/300 mg q.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
  ethinyl estradiol: oral contraceptives formulated with 30-35 μg ethinyl estradiol
- ATV/RTV/TFV 300/100/300mg q.d. With ENG MOTHER: HIV- infected women 2-12 weeks (14-84 days) postpartum who received atazanavir/ritonavir/tenofovir 300/100/300 mg q.d. postpartum and starting postpartum etonogestrel implant atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
  etonogestrel implant: etonogestrel implant contraceptive
- At Least Two 2nd Line TB Drugs w/ or w/Out ARVs INFANT: Infants of HIV-infected and HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following second line TB drugs at study entry:
  Injectable agents:
  * kanamycin
  * amikacin
  * capreomycin
  * Fluoroquinolones:
  * moxifloxacin
  * levofloxacin
  * ofloxacin
  * Oral bacteriostatic second-line agents:
  * ethionamide/prothionamide
  * terizidone/cycloserine
  * para-aminosalicylic acid (PAS)
  * Other agents:
  * high dose INH
  * bedaquiline
  * clofazamine
  * delamanid
  * linezolid
  * pretomanid
- At Least Two 2nd Line TB Drugs w/ or w/Out ARVs MOTHER: HIV-infected and HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following second line TB drugs at study entry:
  Injectable agents:
  * kanamycin
  * amikacin
  * capreomycin
  * Fluoroquinolones:
  * moxifloxacin
  * levofloxacin
  * ofloxacin
  * Oral bacteriostatic second-line agents:
  * ethionamide/prothionamide
  * terizidone/cycloserine
  * para-aminosalicylic acid (PAS)
  * Other agents:
  * high dose INH
  * bedaquiline
  * clofazamine
  * delamanid
  * linezolid
  * pretomanid
- DDI 400mg or 250mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received didanosine delayed release (Videx® EC) 400 mg once a day if weight > 60 kg; 250 mg once a day if weight < 60 kg didanosine delayed release (Videx® EC): didanosine delayed release (Videx® EC) 400 mg once a day if weight > 60 kg; 250 mg once a day if weight < 60 kg
- DDI 400mg or 250mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received didanosine delayed release (Videx® EC) 400 mg once a day if weight > 60 kg; 250 mg once a day if weight < 60 kg didanosine delayed release (Videx® EC): didanosine delayed release (Videx® EC) 400 mg once a day if weight > 60 kg; 250 mg once a day if weight < 60 kg
- DRV/COBI 800/150 mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received darunavir/cobicistat 800/150 mg q.d.
  darunavir/cobicistat: darunavir/cobicistat 800/150 mg q.d.
- DRV/COBI 800/150 mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received darunavir/cobicistat 800/150 mg q.d.
  darunavir/cobicistat: darunavir/cobicistat 800/150 mg q.d.
- DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With 30-35ug EE MOTHER: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received darunavir/cobicistat 800/150 mg q.d. or atazanavir/cobicistat 300/150 mg q.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol atazanavir/cobicistat: atazanavir/cobicistat 300/150 mg q.d. darunavir/cobicistat: darunavir/cobicistat 800/150 mg q.d. ethinyl estradiol: oral contraceptives formulated with 30-35 μg ethinyl estradiol
- DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With ENG MOTHER: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received darunavir/cobicistat 800/150 mg q.d. or atazanavir/cobicistat 300/150 mg q.d. postpartum and starting etonogestrel implant atazanavir/cobicistat: atazanavir/cobicistat 300/150 mg q.d. darunavir/cobicistat: darunavir/cobicistat 800/150 mg q.d. etonogestrel implant: etonogestrel implant contraceptive
- DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received:
  darunavir/ritonavir twice daily 600/100 mg b.i.d. or 800/100 mg b.i.d. until 30 weeks gestation; then 800/100 mg b.i.d. until postpartum hospital discharge; then 600/100 mg b.i.d. after postpartum hospital discharge until 2 week postpartum PK samples are drawn.
  OR darunavir/ritonavir twice daily 600/100 mg b.i.d. or 900/100 mg b.i.d. until 30 weeks gestation; then 900/100 mg b.i.d. until postpartum hospital discharge; then 600/100 mg b.i.d. after postpartum hospital discharge until 2 week postpartum PK samples are drawn.
  darunavir/ritonavir dosage #1: darunavir/ritonavir twice daily 600/100 mg b.i.d.
  darunavir/ritonavir dosage #2: darunavir/ritonavir twice daily 800/100 mg b.i.d.
  darunavir/ritonavir dosage #3: darunavir/ritonavir twice daily 900/100 mg b.i.d.
- DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received:
  darunavir/ritonavir twice daily 600/100 mg b.i.d. or 800/100 mg b.i.d. until 30 weeks gestation; then 800/100 mg b.i.d. until postpartum hospital discharge; then 600/100 mg b.i.d. after postpartum hospital discharge until 2 week postpartum PK samples are drawn.
  OR darunavir/ritonavir twice daily 600/100 mg b.i.d. or 900/100 mg b.i.d. until 30 weeks gestation; then 900/100 mg b.i.d. until postpartum hospital discharge; then 600/100 mg b.i.d. after postpartum hospital discharge until 2 week postpartum PK samples are drawn.
  darunavir/ritonavir dosage #1: darunavir/ritonavir twice daily 600/100 mg b.i.d.
  darunavir/ritonavir dosage #2: darunavir/ritonavir twice daily 800/100 mg b.i.d.
  darunavir/ritonavir dosage #3: darunavir/ritonavir twice daily 900/100 mg b.i.d.
- DRV/RTV 600/100mg b.i.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received darunavir/ritonavir 600/100 mg twice a day darunavir/ritonavir dosage #1: darunavir/ritonavir twice daily 600/100 mg b.i.d.
- DRV/RTV 600/100mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received darunavir/ritonavir 600/100 mg twice a day darunavir/ritonavir dosage #1: darunavir/ritonavir twice daily 600/100 mg b.i.d.
- DRV/RTV 800/100mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received darunavir/ritonavir 800/100 mg once a day darunavir/ritonavir dosage #4: darunavir/ritonavir once daily 800/100 mg q.d.
- DTG 50mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received dolutegravir 50 mg q.d.
  dolutegravir: dolutegravir 50 mg q.d.
- DTG 50mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received dolutegravir 50 mg q.d.
  dolutegravir: dolutegravir 50 mg q.d.
- EFV 600 mg q.d. (Outside THA) INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received efavirenz 600 mg q.d. (Participants outside of Thailand only) efavirenz: efavirenz 600 mg q.d.
- EFV 600 mg q.d. (Outside THA) MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received efavirenz 600 mg q.d. (Participants outside of Thailand only) efavirenz: efavirenz 600 mg q.d.
- EFV 600mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz 600 mg once a day efavirenz: efavirenz 600 mg q.d.
- EFV 600mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz 600 mg once a day efavirenz: efavirenz 600 mg q.d.
- EFV 600mg q.d. and at Least One 1st Line TB Drug INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz 600mg q.d.and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
- EFV 600mg q.d. and at Least One 1st Line TB Drug MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received efavirenz 600mg q.d.and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
- EFV 600mg q.d. With 30-35ug EE MOTHER: HIV-infected women 2-12 weeks (14-84 days) post-delivery who received efavirenz 600mg q.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol efavirenz: efavirenz 600 mg q.d. ethinyl estradiol: oral contraceptives formulated with 30-35 μg ethinyl estradiol
- EFV 600mg q.d. With ENG MOTHER: HIV-infected women 2-12 weeks (14-84 days) postpartum who received efavirenz 600mg q.d. postpartum and starting postpartum etonogestrel implant efavirenz: efavirenz 600 mg q.d. etonogestrel implant: etonogestrel implant contraceptive
- ETR 200mg b.i.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received etravirine 200mg twice a day etravirine: etravirine 200 mg twice a day
- ETR 200mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received etravirine 200mg twice a day etravirine: etravirine 200 mg twice a day
- EVG/COBI 150/150mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received elvitegravir/cobicistat 150/150 mg q.d elvitegravir/cobicistat: elvitegravir/cobicistat 150/150 mg q.d.
- EVG/COBI 150/150mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received elvitegravir/cobicistat 150/150 mg q.d elvitegravir/cobicistat: elvitegravir/cobicistat 150/150 mg q.d.
- FPV/RTV 700/100 b.i.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received fosamprenavir/ritonavir 700/100mg twice a day fosamprenavir/ritonavir: fosamprenavir/ritonavir 700/100 mg twice a day
- FPV/RTV 700/100 b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received fosamprenavir/ritonavir 700/100mg twice a day fosamprenavir/ritonavir: fosamprenavir/ritonavir 700/100 mg twice a day
- FTC 200mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received emtricitabine 200 mg once a day emtricitabine: emtricitabine 200 mg once a day
- FTC 200mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received emtricitabine 200 mg once a day emtricitabine: emtricitabine 200 mg once a day
- IDV/RTV 400/100mg q.d. (Only THA) INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received indinavir/ritonavir 400/100 mg twice a day only to participants enrolling in Thailand indinavir/ritonavir dosage #2: indinavir/ritonavir 400/100 mg twice a day
- IDV/RTV 400/100mg q.d. (Only THA) MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received indinavir/ritonavir 400/100 mg twice a day only to participants enrolling in Thailand indinavir/ritonavir dosage #2: indinavir/ritonavir 400/100 mg twice a day
- IDV/RTV 800/100mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 26 weeks gestation who received indinavir/ritonavir 800/100 mg twice a day indinavir/ritonavir dosage #1: indinavir/ritonavir 800/100mg twice a day
- LPV/RTV 400/100 b.i.d. With 30-35ug EE MOTHER: HIV- infected women 2-12 weeks (14-84 days) postpartum who received lopinavir/ritonavir 400/100 b.i.d. postpartum and starting combined oral contraceptives formulated with 30-35 μg ethinyl estradiol ethinyl estradiol: oral contraceptives formulated with 30-35 μg ethinyl estradiol lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day
- LPV/RTV 400/100 b.i.d. With ENG MOTHER: HIV- infected women 2-12 weeks (14-84 days) postpartum who received lopinavir/ritonavir 400/100 b.i.d. postpartum and starting postpartum etonogestrel implant etonogestrel implant: etonogestrel implant contraceptive lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day
- LPV/RTV 400/100mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 26 weeks gestation who received lopinavir/ritonavir (Kaletra) 400/100mg twice a day lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day
- LPV/RTV 400/100mg b.i.d. Then 533/133mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received Kaletra 400/100 mg twice a day until 30 weeks gestation, then 533/133 mg twice a day until results of postpartum PK evaluation were available lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day lopinavir/ritonavir dosage #3: lopinavir/ritonavir (Kaletra) 533/133 mg twice a day
- LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites) INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir (Alluvia tablets) 400/100 mg [2 tablets] twice day until 30 weeks gestation; then 600/150 mg [3 tablets] twice a day until postpartum hospital discharge; then 400/100 mg [2 tablets] twice a day after postpartum hospital discharge until 2 week postpartum PK sample drawn only to participants enrolling in Uganda lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day lopinavir/ritonavir dosage #4: lopinavir/ritonavir (Kaletra) tablets 600/150 mg [3 tablets] twice a day
- LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites) MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir (Alluvia tablets) 400/100 mg [2 tablets] twice day until 30 weeks gestation; then 600/150 mg [3 tablets] twice a day until postpartum hospital discharge; then 400/100 mg [2 tablets] twice a day after postpartum hospital discharge until 2 week postpartum PK sample drawn only to participants enrolling in Uganda lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day lopinavir/ritonavir dosage #4: lopinavir/ritonavir (Kaletra) tablets 600/150 mg [3 tablets] twice a day
- LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir (Kaletra) tablets 400/100 mg [2 tablets] twice a day until 30 weeks gestation, then 600/150 mg [3 tablets] twice a day until postpartum hospital discharge; and 400/100 mg [2 tablets] twice a day after postpartum hospital discharge, until 2 week postpartum PK sample is drawn lopinavir/ritonavir dosage #2: lopinavir/ritonavir (Kaletra) 400/100mg twice a day lopinavir/ritonavir dosage #4: lopinavir/ritonavir (Kaletra) tablets 600/150 mg [3 tablets] twice a day
- LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir 800/200mg b.i.d. and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
- LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received lopinavir/ritonavir 800/200mg b.i.d. and TB treatment with at least one of the following TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
- MVC 150 or 300mg b.i.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received maraviroc 150 mg or 300 mg twice a day maraviroc: maraviroc 150 mg or 300 mg twice a day
- MVC 150 or 300mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received maraviroc 150 mg or 300 mg twice a day maraviroc: maraviroc 150 mg or 300 mg twice a day
- NFV 1250mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received nelfinavir [625 mg tablets] 1250 mg twice a day nelfinavir dosage #1: nelfinavir [625 mg tablets] 1250 mg twice a day
- NFV 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received nelfinavir [625 mg tablets] 1250 mg twice a day until 30 weeks gestation; then 1875 mg twice a day until postpartum hospital discharge; then 1250 mg twice a day after postpartum hospital discharge until 2 week postpartum PK samples drawn nelfinavir dosage #1: nelfinavir [625 mg tablets] 1250 mg twice a day nelfinavir dosage #2: nelfinavir [625 mg tablets] 1875 mg twice a day
- NVP 200mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 26 weeks gestation who received nevirapine 200 mg twice a day nevirapine: nevirapine 200 mg twice a day
- No ARVs and at Least Two 1st Line TB Drugs INFANT: Infants of HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following first line TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
- No ARVs and at Least Two 1st Line TB Drugs MOTHER: HIV-uninfected pregnant women ≥ 20 weeks gestation who received at least two of the following first line TB drugs at study entry:
  * rifampicin 8-12 mg/kg (max 600 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * ethambutol 15-20 mg/kg q.d., 25-35 mg/kg t.i.w.
  * isoniazid 4-6 mg/kg (max 300 mg) q.d.; 8-12 mg/kg (max 900 mg) t.i.w.
  * pyrazinamide 20-30mg/kg q.d.; 30-40mg/kg t.i.w.
- RAL 400mg b.i.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received raltegravir 400 mg twice a day raltegravir: raltegravir 400 mg twice a day
- RAL 400mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received raltegravir 400 mg twice a day raltegravir: raltegravir 400 mg twice a day
- RPV 25mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received rilpivirine (25 mg q.d.) rilpivirine: rilpivirine (25 mg q.d.)
- RPV 25mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received rilpivirine (25 mg q.d.) rilpivirine: rilpivirine (25 mg q.d.)
- TAF 10mg q.d. w/COBI INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 10 mg q.d. with cobicistat.
  TAF w/cobicistat: TAF 10 mg q.d. with cobicistat
- TAF 10mg q.d. w/COBI MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 10 mg q.d. with cobicistat.
  TAF w/cobicistat: TAF 10 mg q.d. with cobicistat
- TAF 25mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 25 mg q.d. without cobicistat or ritonavir boosting.
  tenofovir alafenamide fumarate (TAF): TAF 25 mg q.d. without cobicistat or ritonavir boosting
- TAF 25mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 25 mg q.d. without cobicistat or ritonavir boosting.
  tenofovir alafenamide fumarate (TAF): TAF 25 mg q.d. without cobicistat or ritonavir boosting
- TAF 25mg q.d. w/COBI or RTV Boosting INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 25 mg q.d. with cobicistat or ritonavir boosting.
  TAF w/cobicistat or ritonavir: TAF 25 mg q.d. with cobicistat or ritonavir boosting
- TAF 25mg q.d. w/COBI or RTV Boosting MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation NOT on tuberculosis treatment who received tenofovir alafenamide fumarate (TAF) 25 mg q.d. with cobicistat or ritonavir boosting.
  TAF w/cobicistat or ritonavir: TAF 25 mg q.d. with cobicistat or ritonavir boosting
- TFV 300mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir 300 mg once a day tenofovir: tenofovir 300 mg once a day
- TFV/ATV/RTV 300/300/100mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir/atazanavir/ritonavir 300/300/100 mg once a day atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
- TFV/ATV/RTV 300/300/100mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir/atazanavir/ritonavir 300/300/100 mg once a day atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
- TFV/ATV/RTV 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. INFANT: Infants of HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir/atazanavir/ritonavir 300/300/100 mg once a day until 30 weeks gestation; then 300/400/100 mg once a day until postpartum hospital discharge; then 300/300/100 mg once a day after postpartum hospital discharge until 2 week postpartum PK samples drawn atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
  tenofovir/atazanavir/ritonavir dosage #2: tenofovir/atazanavir/ritonavir 300/400/100 mg once a day
- TFV/ATV/RTV 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received tenofovir/atazanavir/ritonavir 300/300/100 mg once a day until 30 weeks gestation; then 300/400/100 mg once a day until postpartum hospital discharge; then 300/300/100 mg once a day after postpartum hospital discharge until 2 week postpartum PK samples drawn atazanavir/ritonavir/tenofovir dosage #1: atazanavir/ritonavir/tenofovir 300/100/300mg q.d.
  tenofovir/atazanavir/ritonavir dosage #2: tenofovir/atazanavir/ritonavir 300/400/100 mg once a day
- TPV/RTV 500/200mg b.i.d. MOTHER: HIV-infected pregnant women ≥ 20 weeks gestation who received tipranavir/ritonavir (TPV/RTV) 500/200 mg twice a day
  tipranavir/ritonavir: tipranavir/ritonavir 500/200 mg twice a day
Arm/Group | ABC 300mg b.i.d. MOTHER | ATV/COBI 300/150 mg q.d. INFANT | ATV/COBI 300/150 mg q.d. MOTHER | ATV/RTV 300/100mg q.d. INFANT | ATV/RTV 300/100mg q.d. MOTHER | ATV/RTV 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. INFANT | ATV/RTV 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. MOTHER | ATV/RTV/TFV 300/100/300mg q.d. With 30-35ug EE MOTHER | ATV/RTV/TFV 300/100/300mg q.d. With ENG MOTHER | At Least Two 2nd Line TB Drugs w/ or w/Out ARVs INFANT | At Least Two 2nd Line TB Drugs w/ or w/Out ARVs MOTHER | DDI 400mg or 250mg q.d. INFANT | DDI 400mg or 250mg q.d. MOTHER | DRV/COBI 800/150 mg q.d. INFANT | DRV/COBI 800/150 mg q.d. MOTHER | DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With 30-35ug EE MOTHER | DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With ENG MOTHER | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. INFANT | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. MOTHER | DRV/RTV 600/100mg b.i.d. INFANT | DRV/RTV 600/100mg b.i.d. MOTHER | DRV/RTV 800/100mg q.d. MOTHER | DTG 50mg q.d. INFANT | DTG 50mg q.d. MOTHER | EFV 600 mg q.d. (Outside THA) INFANT | EFV 600 mg q.d. (Outside THA) MOTHER | EFV 600mg q.d. INFANT | EFV 600mg q.d. MOTHER | EFV 600mg q.d. and at Least One 1st Line TB Drug INFANT | EFV 600mg q.d. and at Least One 1st Line TB Drug MOTHER | EFV 600mg q.d. With 30-35ug EE MOTHER | EFV 600mg q.d. With ENG MOTHER | ETR 200mg b.i.d. INFANT | ETR 200mg b.i.d. MOTHER | EVG/COBI 150/150mg q.d. INFANT | EVG/COBI 150/150mg q.d. MOTHER | FPV/RTV 700/100 b.i.d. INFANT | FPV/RTV 700/100 b.i.d. MOTHER | FTC 200mg q.d. INFANT | FTC 200mg q.d. MOTHER | IDV/RTV 400/100mg q.d. (Only THA) INFANT | IDV/RTV 400/100mg q.d. (Only THA) MOTHER | IDV/RTV 800/100mg b.i.d. MOTHER | LPV/RTV 400/100 b.i.d. With 30-35ug EE MOTHER | LPV/RTV 400/100 b.i.d. With ENG MOTHER | LPV/RTV 400/100mg b.i.d. MOTHER | LPV/RTV 400/100mg b.i.d. Then 533/133mg b.i.d. MOTHER | LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites) INFANT | LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites) MOTHER | LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. MOTHER | LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug INFANT | LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug MOTHER | MVC 150 or 300mg b.i.d. INFANT | MVC 150 or 300mg b.i.d. MOTHER | NFV 1250mg b.i.d. MOTHER | NFV 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d. MOTHER | NVP 200mg b.i.d. MOTHER | No ARVs and at Least Two 1st Line TB Drugs INFANT | No ARVs and at Least Two 1st Line TB Drugs MOTHER | RAL 400mg b.i.d. INFANT | RAL 400mg b.i.d. MOTHER | RPV 25mg q.d. INFANT | RPV 25mg q.d. MOTHER | TAF 10mg q.d. w/COBI INFANT | TAF 10mg q.d. w/COBI MOTHER | TAF 25mg q.d. INFANT | TAF 25mg q.d. MOTHER | TAF 25mg q.d. w/COBI or RTV Boosting INFANT | TAF 25mg q.d. w/COBI or RTV Boosting MOTHER | TFV 300mg q.d. MOTHER | TFV/ATV/RTV 300/300/100mg q.d. INFANT | TFV/ATV/RTV 300/300/100mg q.d. MOTHER | TFV/ATV/RTV 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. INFANT | TFV/ATV/RTV 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. MOTHER | TPV/RTV 500/200mg b.i.d. MOTHER
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/12 | 0/12 | 0/22 | 0/22 | 0/38 | 0/38 | 0/28 | 0/25 | 0/14 | 0/13 | 0/4 | 0/18 | 0/27 | 0/28 | 0/2 | 0/6 | 0/25 | 0/26 | 1/9 | 0/36 | 0/32 | 0/30 | 0/30 | 0/26 | 0/27 | 0/21 | 0/25 | 1/23 | 0/24 | 0/29 | 0/28 | 0/6 | 0/16 | 0/31 | 0/31 | 0/9 | 0/30 | 0/5 | 0/21 | 0/26 | 0/26 | 0/1 | 0/27 | 0/27 | 0/17 | 0/29 | 1/25 | 0/25 | 0/35 | 0/2 | 0/2 | 0/4 | 0/12 | 0/29 | 0/18 | 0/12 | 2/27 | 0/27 | 0/6 | 0/43 | 0/30 | 0/32 | 0/32 | 0/33 | 0/27 | 0/27 | 0/28 | 0/29 | 0/28 | 0/21 | 0/25 | 0/35 | 0/35 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/26 | 3/12 | 3/12 | 0/22 | 1/22 | 6/38 | 0/38 | 2/28 | 0/25 | 8/14 | 4/13 | 0/4 | 0/18 | 7/27 | 5/28 | 0/2 | 0/6 | 0/25 | 3/26 | 1/9 | 0/36 | 0/32 | 7/30 | 3/30 | 8/26 | 5/27 | 0/21 | 0/25 | 7/23 | 6/24 | 3/29 | 0/28 | 1/6 | 1/16 | 5/31 | 5/31 | 2/9 | 0/30 | 0/5 | 1/21 | 0/26 | 0/26 | 0/1 | 0/27 | 0/27 | 0/17 | 0/29 | 3/25 | 3/25 | 1/35 | 2/2 | 0/2 | 0/4 | 0/12 | 0/29 | 2/18 | 0/12 | 7/27 | 6/27 | 1/6 | 0/43 | 3/30 | 2/32 | 10/32 | 7/33 | 4/27 | 4/27 | 5/28 | 5/29 | 0/28 | 2/21 | 1/25 | 2/35 | 0/35 | 0/1
Other Adverse Events (participants affected / at risk) | 21/26 | 9/12 | 11/12 | 8/22 | 21/22 | 23/38 | 36/38 | 27/28 | 19/25 | 8/14 | 12/13 | 2/4 | 14/18 | 18/27 | 23/28 | 1/2 | 4/6 | 22/25 | 24/26 | 5/9 | 28/36 | 29/32 | 25/30 | 29/30 | 16/26 | 27/27 | 11/21 | 24/25 | 14/23 | 23/24 | 21/29 | 21/28 | 4/6 | 16/16 | 17/31 | 26/31 | 8/9 | 28/30 | 2/5 | 18/21 | 11/26 | 25/26 | 1/1 | 16/27 | 17/27 | 13/17 | 28/29 | 12/25 | 25/25 | 34/35 | 2/2 | 2/2 | 3/4 | 9/12 | 21/29 | 17/18 | 9/12 | 16/27 | 27/27 | 3/6 | 40/43 | 24/30 | 30/32 | 24/32 | 30/33 | 20/27 | 23/27 | 18/28 | 27/29 | 21/28 | 11/21 | 24/25 | 16/35 | 35/35 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABC 300mg b.i.d. MOTHER (N=26) | ATV/COBI 300/150 mg q.d. INFANT (N=12) | ATV/COBI 300/150 mg q.d. MOTHER (N=12) | ATV/RTV 300/100mg q.d. INFANT (N=22) | ATV/RTV 300/100mg q.d. MOTHER (N=22) | ATV/RTV 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. INFANT (N=38) | ATV/RTV 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. MOTHER (N=38) | ATV/RTV/TFV 300/100/300mg q.d. With 30-35ug EE MOTHER (N=28) | ATV/RTV/TFV 300/100/300mg q.d. With ENG MOTHER (N=25) | At Least Two 2nd Line TB Drugs w/ or w/Out ARVs INFANT (N=14) | At Least Two 2nd Line TB Drugs w/ or w/Out ARVs MOTHER (N=13) | DDI 400mg or 250mg q.d. INFANT (N=4) | DDI 400mg or 250mg q.d. MOTHER (N=18) | DRV/COBI 800/150 mg q.d. INFANT (N=27) | DRV/COBI 800/150 mg q.d. MOTHER (N=28) | DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With 30-35ug EE MOTHER (N=2) | DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With ENG MOTHER (N=6) | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. INFANT (N=25) | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. MOTHER (N=26) | DRV/RTV 600/100mg b.i.d. INFANT (N=9) | DRV/RTV 600/100mg b.i.d. MOTHER (N=36) | DRV/RTV 800/100mg q.d. MOTHER (N=32) | DTG 50mg q.d. INFANT (N=30) | DTG 50mg q.d. MOTHER (N=30) | EFV 600 mg q.d. (Outside THA) INFANT (N=26) | EFV 600 mg q.d. (Outside THA) MOTHER (N=27) | EFV 600mg q.d. INFANT (N=21) | EFV 600mg q.d. MOTHER (N=25) | EFV 600mg q.d. and at Least One 1st Line TB Drug INFANT (N=23) | EFV 600mg q.d. and at Least One 1st Line TB Drug MOTHER (N=24) | EFV 600mg q.d. With 30-35ug EE MOTHER (N=29) | EFV 600mg q.d. With ENG MOTHER (N=28) | ETR 200mg b.i.d. INFANT (N=6) | ETR 200mg b.i.d. MOTHER (N=16) | EVG/COBI 150/150mg q.d. INFANT (N=31) | EVG/COBI 150/150mg q.d. MOTHER (N=31) | FPV/RTV 700/100 b.i.d. INFANT (N=9) | FPV/RTV 700/100 b.i.d. MOTHER (N=30) | FTC 200mg q.d. INFANT (N=5) | FTC 200mg q.d. MOTHER (N=21) | IDV/RTV 400/100mg q.d. (Only THA) INFANT (N=26) | IDV/RTV 400/100mg q.d. (Only THA) MOTHER (N=26) | IDV/RTV 800/100mg b.i.d. MOTHER (N=1) | LPV/RTV 400/100 b.i.d. With 30-35ug EE MOTHER (N=27) | LPV/RTV 400/100 b.i.d. With ENG MOTHER (N=27) | LPV/RTV 400/100mg b.i.d. MOTHER (N=17) | LPV/RTV 400/100mg b.i.d. Then 533/133mg b.i.d. MOTHER (N=29) | LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites) INFANT (N=25) | LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites) MOTHER (N=25) | LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. MOTHER (N=35) | LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug INFANT (N=2) | LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug MOTHER (N=2) | MVC 150 or 300mg b.i.d. INFANT (N=4) | MVC 150 or 300mg b.i.d. MOTHER (N=12) | NFV 1250mg b.i.d. MOTHER (N=29) | NFV 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d. MOTHER (N=18) | NVP 200mg b.i.d. MOTHER (N=12) | No ARVs and at Least Two 1st Line TB Drugs INFANT (N=27) | No ARVs and at Least Two 1st Line TB Drugs MOTHER (N=27) | RAL 400mg b.i.d. INFANT (N=6) | RAL 400mg b.i.d. MOTHER (N=43) | RPV 25mg q.d. INFANT (N=30) | RPV 25mg q.d. MOTHER (N=32) | TAF 10mg q.d. w/COBI INFANT (N=32) | TAF 10mg q.d. w/COBI MOTHER (N=33) | TAF 25mg q.d. INFANT (N=27) | TAF 25mg q.d. MOTHER (N=27) | TAF 25mg q.d. w/COBI or RTV Boosting INFANT (N=28) | TAF 25mg q.d. w/COBI or RTV Boosting MOTHER (N=29) | TFV 300mg q.d. MOTHER (N=28) | TFV/ATV/RTV 300/300/100mg q.d. INFANT (N=21) | TFV/ATV/RTV 300/300/100mg q.d. MOTHER (N=25) | TFV/ATV/RTV 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. INFANT (N=35) | TFV/ATV/RTV 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. MOTHER (N=35) | TPV/RTV 500/200mg b.i.d. MOTHER (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anomalous pulmonary venous connection (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asphyxiating thoracic dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital anaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital naevus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Congenital pseudarthrosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital syphilis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmorphism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypospadias (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney duplex (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngomalacia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polydactyly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infantile spitting up (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug withdrawal syndrome neonatal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden infant death syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis of pregnancy (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis fulminant (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HIV test (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza A virus test (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intra-abdominal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure like phenomena (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonic posturing (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foetal cardiac disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peyronie's disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABC 300mg b.i.d. MOTHER (N=26) | ATV/COBI 300/150 mg q.d. INFANT (N=12) | ATV/COBI 300/150 mg q.d. MOTHER (N=12) | ATV/RTV 300/100mg q.d. INFANT (N=22) | ATV/RTV 300/100mg q.d. MOTHER (N=22) | ATV/RTV 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. INFANT (N=38) | ATV/RTV 300/100mg q.d. Then 400/100mg q.d. Then 300/100mg q.d. MOTHER (N=38) | ATV/RTV/TFV 300/100/300mg q.d. With 30-35ug EE MOTHER (N=28) | ATV/RTV/TFV 300/100/300mg q.d. With ENG MOTHER (N=25) | At Least Two 2nd Line TB Drugs w/ or w/Out ARVs INFANT (N=14) | At Least Two 2nd Line TB Drugs w/ or w/Out ARVs MOTHER (N=13) | DDI 400mg or 250mg q.d. INFANT (N=4) | DDI 400mg or 250mg q.d. MOTHER (N=18) | DRV/COBI 800/150 mg q.d. INFANT (N=27) | DRV/COBI 800/150 mg q.d. MOTHER (N=28) | DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With 30-35ug EE MOTHER (N=2) | DRV/COBI 800/150mg q.d. or ATV/COBI 300/150mg q.d With ENG MOTHER (N=6) | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. INFANT (N=25) | DRV/RTV 600 or 800 or 900/100mg b.i.d. Then 800 or 900/100mg b.i.d. Then 600/100mg b.i.d. MOTHER (N=26) | DRV/RTV 600/100mg b.i.d. INFANT (N=9) | DRV/RTV 600/100mg b.i.d. MOTHER (N=36) | DRV/RTV 800/100mg q.d. MOTHER (N=32) | DTG 50mg q.d. INFANT (N=30) | DTG 50mg q.d. MOTHER (N=30) | EFV 600 mg q.d. (Outside THA) INFANT (N=26) | EFV 600 mg q.d. (Outside THA) MOTHER (N=27) | EFV 600mg q.d. INFANT (N=21) | EFV 600mg q.d. MOTHER (N=25) | EFV 600mg q.d. and at Least One 1st Line TB Drug INFANT (N=23) | EFV 600mg q.d. and at Least One 1st Line TB Drug MOTHER (N=24) | EFV 600mg q.d. With 30-35ug EE MOTHER (N=29) | EFV 600mg q.d. With ENG MOTHER (N=28) | ETR 200mg b.i.d. INFANT (N=6) | ETR 200mg b.i.d. MOTHER (N=16) | EVG/COBI 150/150mg q.d. INFANT (N=31) | EVG/COBI 150/150mg q.d. MOTHER (N=31) | FPV/RTV 700/100 b.i.d. INFANT (N=9) | FPV/RTV 700/100 b.i.d. MOTHER (N=30) | FTC 200mg q.d. INFANT (N=5) | FTC 200mg q.d. MOTHER (N=21) | IDV/RTV 400/100mg q.d. (Only THA) INFANT (N=26) | IDV/RTV 400/100mg q.d. (Only THA) MOTHER (N=26) | IDV/RTV 800/100mg b.i.d. MOTHER (N=1) | LPV/RTV 400/100 b.i.d. With 30-35ug EE MOTHER (N=27) | LPV/RTV 400/100 b.i.d. With ENG MOTHER (N=27) | LPV/RTV 400/100mg b.i.d. MOTHER (N=17) | LPV/RTV 400/100mg b.i.d. Then 533/133mg b.i.d. MOTHER (N=29) | LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites) INFANT (N=25) | LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. (Only African Sites) MOTHER (N=25) | LPV/RTV 400/100mg b.i.d. Then 600/150mg b.i.d. Then 400/100mg b.i.d. MOTHER (N=35) | LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug INFANT (N=2) | LPV/RTV 800/200mg b.i.d. and at Least One 1st Line TB Drug MOTHER (N=2) | MVC 150 or 300mg b.i.d. INFANT (N=4) | MVC 150 or 300mg b.i.d. MOTHER (N=12) | NFV 1250mg b.i.d. MOTHER (N=29) | NFV 1250mg b.i.d. Then 1875mg b.i.d. Then 1250mg b.i.d. MOTHER (N=18) | NVP 200mg b.i.d. MOTHER (N=12) | No ARVs and at Least Two 1st Line TB Drugs INFANT (N=27) | No ARVs and at Least Two 1st Line TB Drugs MOTHER (N=27) | RAL 400mg b.i.d. INFANT (N=6) | RAL 400mg b.i.d. MOTHER (N=43) | RPV 25mg q.d. INFANT (N=30) | RPV 25mg q.d. MOTHER (N=32) | TAF 10mg q.d. w/COBI INFANT (N=32) | TAF 10mg q.d. w/COBI MOTHER (N=33) | TAF 25mg q.d. INFANT (N=27) | TAF 25mg q.d. MOTHER (N=27) | TAF 25mg q.d. w/COBI or RTV Boosting INFANT (N=28) | TAF 25mg q.d. w/COBI or RTV Boosting MOTHER (N=29) | TFV 300mg q.d. MOTHER (N=28) | TFV/ATV/RTV 300/300/100mg q.d. INFANT (N=21) | TFV/ATV/RTV 300/300/100mg q.d. MOTHER (N=25) | TFV/ATV/RTV 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. INFANT (N=35) | TFV/ATV/RTV 300/300/100mg q.d. Then 300/400/100mg q.d Then 300/300/100mg q.d. MOTHER (N=35) | TPV/RTV 500/200mg b.i.d. MOTHER (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia neonatal (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect acquired (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
ABO haemolytic disease of newborn (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital HIV infection (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital central nervous system anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital choroid plexus cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital genital malformation female (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital musculoskeletal anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital naevus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital toxoplasmosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Craniotabes (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sickle cell trait (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Conjunctival discolouration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival pallor (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 3 | 3 | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 1 | 3 | 0 | 3 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 6 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 1 | 3 | 1 | 4 | 0 | 1 | 2 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 3 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 4 | 0 | 2 | 0
Adverse event (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 0 | 2 | 3 | 3 | 1 | 4 | 2 | 2 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 2 | 1 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis of pregnancy (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 0
Immunisation reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amniotic cavity infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 4 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cervicitis human papilloma virus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cervicitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometritis decidual (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis neonatal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vaginitis gardnerella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vulvovaginitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginitis trichomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 5 | 0 | 3 | 4 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 4 | 8 | 0 | 3 | 0 | 5 | 0 | 4 | 0 | 5 | 5 | 6 | 0 | 4 | 1 | 3 | 1 | 8 | 0 | 3 | 0 | 1 | 0 | 1 | 2 | 1 | 4 | 0 | 2 | 5 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 6 | 0 | 8 | 0 | 7 | 0 | 0 | 1 | 1 | 0 | 3 | 4 | 0 | 4 | 0 | 6 | 0
Amylase increased (Investigations) | 3 | 0 | 0 | 0 | 9 | 0 | 13 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 1 | 6 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 5 | 0 | 6 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 2 | 1 | 2 | 5 | 4 | 5 | 1 | 0 | 3 | 0 | 3 | 3 | 1 | 1 | 0 | 0 | 5 | 0 | 4 | 8 | 4 | 7 | 0 | 4 | 0 | 5 | 1 | 7 | 3 | 5 | 0 | 3 | 2 | 5 | 2 | 10 | 0 | 4 | 1 | 3 | 0 | 1 | 0 | 2 | 4 | 0 | 2 | 10 | 0 | 0 | 0 | 2 | 3 | 1 | 2 | 1 | 8 | 1 | 7 | 0 | 9 | 1 | 2 | 1 | 4 | 2 | 2 | 5 | 1 | 4 | 2 | 5 | 0
Bilirubin conjugated increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 9 | 0 | 0 | 2 | 15 | 0 | 0 | 1 | 7 | 0 | 0 | 0 | 1 | 21 | 0 | 17 | 0 | 0 | 0 | 20 | 1 | 0 | 1 | 6 | 1 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 1 | 15 | 0 | 13 | 0 | 12 | 0 | 13 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 6 | 0 | 2 | 0 | 10 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 7 | 0 | 4 | 0 | 2 | 2 | 9 | 0 | 4 | 8 | 0 | 2 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 9 | 0 | 10 | 0 | 3 | 1 | 0 | 0 | 2 | 12 | 0 | 0 | 18 | 0 | 0 | 0 | 0 | 3 | 10 | 2 | 1 | 2 | 0 | 12 | 1 | 10 | 1 | 1 | 0 | 2 | 0 | 5 | 11 | 0 | 12 | 0 | 17 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 1 | 4 | 15 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 9 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 10 | 0 | 3 | 0 | 4 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 4 | 3 | 4 | 3 | 18 | 2 | 33 | 17 | 13 | 0 | 0 | 0 | 2 | 5 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 8 | 1 | 12 | 0 | 1 | 2 | 3 | 8 | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 3 | 2 | 2 | 18 | 2 | 27 | 0
Blood calcium decreased (Investigations) | 9 | 0 | 2 | 0 | 6 | 0 | 4 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 5 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 1 | 2 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 7 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 15 | 0 | 0 | 13 | 0 | 0 | 0 | 0 | 4 | 4 | 5 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 9 | 0 | 12 | 0 | 12 | 1
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood glucose abnormal (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0 | 5 | 1
Blood glucose decreased (Investigations) | 3 | 3 | 0 | 0 | 10 | 4 | 16 | 2 | 1 | 0 | 0 | 0 | 2 | 2 | 6 | 0 | 0 | 5 | 8 | 0 | 3 | 2 | 10 | 1 | 2 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 3 | 3 | 0 | 3 | 0 | 6 | 2 | 1 | 0 | 0 | 2 | 1 | 13 | 0 | 13 | 13 | 0 | 1 | 0 | 0 | 7 | 10 | 1 | 2 | 0 | 0 | 6 | 4 | 3 | 4 | 0 | 7 | 4 | 2 | 3 | 6 | 0 | 8 | 3 | 16 | 0
Blood glucose increased (Investigations) | 3 | 0 | 1 | 0 | 7 | 0 | 9 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 4 | 0 | 1 | 1 | 2 | 1 | 1 | 9 | 0 | 6 | 15 | 0 | 0 | 0 | 0 | 2 | 4 | 2 | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 2 | 1 | 1 | 0 | 1 | 3 | 0 | 5 | 0 | 6 | 0
Blood magnesium decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 3 | 0 | 0 | 0 | 2 | 1 | 11 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 2 | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 4 | 0 | 0 | 0 | 2 | 0 | 2 | 8 | 0 | 9 | 11 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 8 | 0 | 12 | 1
Blood potassium increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 6 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 10 | 0 | 2 | 0 | 12 | 0 | 20 | 3 | 1 | 0 | 1 | 0 | 5 | 2 | 5 | 0 | 0 | 2 | 14 | 1 | 12 | 10 | 2 | 2 | 0 | 1 | 0 | 2 | 0 | 3 | 3 | 7 | 0 | 3 | 1 | 2 | 0 | 14 | 0 | 11 | 1 | 2 | 1 | 0 | 3 | 7 | 23 | 0 | 22 | 30 | 0 | 1 | 0 | 1 | 12 | 10 | 4 | 1 | 0 | 0 | 12 | 2 | 8 | 0 | 2 | 0 | 0 | 0 | 2 | 16 | 0 | 18 | 1 | 25 | 1
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose tolerance test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 6 | 2 | 3 | 0 | 5 | 9 | 7 | 2 | 5 | 0 | 8 | 0 | 1 | 3 | 14 | 0 | 0 | 6 | 8 | 1 | 9 | 9 | 3 | 11 | 1 | 15 | 4 | 7 | 0 | 15 | 3 | 2 | 2 | 7 | 2 | 11 | 1 | 5 | 0 | 2 | 3 | 8 | 0 | 2 | 0 | 2 | 4 | 5 | 11 | 6 | 0 | 1 | 1 | 6 | 1 | 4 | 3 | 0 | 10 | 2 | 11 | 5 | 12 | 2 | 12 | 0 | 13 | 1 | 15 | 6 | 0 | 4 | 1 | 5 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 0 | 2 | 2 | 4 | 4 | 3 | 2 | 2 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 4 | 2 | 1 | 2 | 0 | 0 | 4 | 3 | 0 | 4 | 2 | 1 | 2 | 3 | 6 | 5 | 0 | 0 | 1 | 1 | 4 | 1 | 4 | 1 | 1 | 0 | 1 | 8 | 1 | 2 | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 2 | 2 | 7 | 0
Platelet count decreased (Investigations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Streptococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Late metabolic acidosis of newborn (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0
Cranial sutures widening (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia neonatal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 6 | 2 | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 6 | 0 | 1 | 0 | 5 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 5 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 6 | 0 | 8 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neonatal seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system cyst (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 1 | 0 | 14 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 6 | 0 | 0
Labour pain (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Maternal condition affecting foetus (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 4 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 6 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine atony (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine hypertonus (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perinatal depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast engorgement (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 0
Cervix inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Shortened cervix (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 5 | 0 | 4 | 6 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 6 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Vulval disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vulval ulceration (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 3 | 1 | 2 | 1 | 4 | 0 | 5 | 2 | 0 | 2 | 4 | 4 | 0 | 1 | 1 | 1 | 0 | 2 | 3 | 3 | 0 | 1 | 3 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 4 | 3 | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 5 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Grunting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 2 | 1 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 2 | 0
Nasal flaring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 0
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neonatal hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Over the course of the study, some study arms were discontinued or closed for reasons such as there being sufficient pharmacokinetic data from other studies or lack of enrollment (as specified in Protocol Section 8.42), leading to a low number of participants in those arms. In addition, due to the COVID-19 pandemic there was a delay in running assays for certain arms and/or analyzing PK results; the results for those arms will be reported when available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (6):
  • Study Protocol: P1026s Protocol Version 10.0_02Feb2016 (2016-02-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT00042289/Prot_001.pdf
  • Study Protocol: P1026s Protocol Version 10.0_Letter of Amendment 1_14Dec2016 (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT00042289/Prot_002.pdf
  • Study Protocol: P1026s Protocol Version 10.0_Letter of Amendment 2_13Apr2018 (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT00042289/Prot_003.pdf
  • Statistical Analysis Plan: PK SAP (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT00042289/SAP_004.pdf
  • Statistical Analysis Plan: Primary SAP (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT00042289/SAP_005.pdf
  • Informed Consent Form (2016-02-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT00042289/ICF_000.pdf